CLINICAL TRIAL: NCT01969344
Title: Subpopulations and Intermediate Outcome Measures in COPD Study
Brief Title: Study of COPD Subgroups and Biomarkers
Acronym: SPIROMICS
Status: Active, not recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); COPD Foundation (Other); Columbia University (Other); Johns Hopkins University (Other); National Jewish Health (Other); Temple University (Other); University of Alabama at Birmingham (Other); University of California, Los Angeles (Other); University of California, San Francisco (Other); University of Illinois at Chicago (Other); University of Iowa (Other); University of Michigan (Other); University of Utah (Other); Wake Forest University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0048; 5U01HL137880 (NIH); 1U24HL141762 (NIH); R01HL144718 (NIH); R01HL093081 (NIH); HHSN268200900020C (Other: National Heart, Lung, and Blood Institute); HHSN268200900013C (Other: National Heart, Lung, and Blood Institute); HHSN268200900014C (Other: National Heart, Lung, and Blood Institute); HHSN268200900015C (Other: National Heart, Lung, and Blood Institute); HHSN268200900016C (Other: National Heart, Lung, and Blood Institute); HHSN268200900017C (Other: National Heart, Lung, and Blood Institute); HHSN268200900018C (Other: National Heart, Lung, and Blood Institute); HHSN2682009000019C (Other: National Heart, Lung, and Blood Institute); 75N92024D00012 (Other: National Heart, Lung, and Blood Institute)
Record Dates: First submitted 2013-10-16; First posted 2013-10-25 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-09

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, urine, lung biopsies, lung bronchial wash and lavage fluid, oral rinse and tongue scrapping, and sputum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Smokers without COPD: Current or former smokers with at least a 20 pack-year history with normal lung function based on post-bronchodilator spirometry (n=944).
- Severe COPD: Current and former smokers with at least a 20 pack-year history with severe COPD based on post-bronchodilator spirometry (n=625).
- Mild/Moderate COPD: Current and former smokers with at least a 20 pack-year history with mild to moderate COPD based on post-bronchodilator spirometry (n=1210).
- Non-smokers: Never-smokers with normal lung function on spirometry without use of bronchodilators (n=201).

SUMMARY:
SPIROMICS I, SPIROMICS II, and SPIROMICS III are longitudinal observational studies of Chronic Obstructive Pulmonary Disease (COPD) cohort.

SPIROMICS I had two primary aims: (1) To find groups of patients with COPD who share certain characteristics; (2) To find new ways of measuring whether or not COPD is getting worse and to provide new ways of testing whether a new treatment is working.

SPIROMICS II had three primary aims: (1) To define the natural history of "smokers with symptoms despite preserved spirometry" and characterize the airway mucus abnormalities underlying this condition; (2) To determine the radiographic precursor lesion(s) for emphysema and identify the molecular phenotypes underlying airway disease and emphysema; (3) To advance understanding of the biology of COPD exacerbations through analysis of predisposing baseline phenotypes, exacerbation triggers and host inflammatory response.

SPIROMICS III has three primary aims: (1) To identify the main forms of smoking-related airway disease that are caused by pathological airway mucus, their biological underpinnings, and their physiological significance; (2) To identify longitudinal trajectories in established and novel CT measures of emphysema, test how they predict COPD progression, and define their underlying biology; (3) To identify environmental and social determinants of health that impact disease severity and progression and their influence on lung structure, biology, and health disparities in COPD.

DETAILED DESCRIPTION:
SPIROMICS was initially funded through contracts from the NIH. That phase of SPIROMICS is now referred to as SPIROMICS I. SPIROMICS II was funded as a grant from the NIH to continue the longitudinal observation of the SPIROMICS cohort recruited in SPIROMICS I. The current phase, referred to as SPIROMICS III, is funded through a contract from the NIH to continue the longitudinal observation of the SPIROMICS cohort that remain active (not withdrawn, lost to follow-up, or deceased).

Description of SPIROMICS I:

The purpose of SPIROMICS was to learn about chronic obstructive pulmonary disease (COPD), which is sometimes called emphysema or chronic bronchitis. Millions of Americans have COPD, and it is the fourth leading cause of death in the country. The most common cause of COPD is cigarette smoking, although not all smokers get COPD. The discovery of new treatments for COPD has been slowed by a poor understanding of different types of COPD and a lack of ways to measure whether or not COPD is getting worse.

The study had two main goals. The first was to find groups of patients with COPD who share certain characteristics. Certain groups may respond differently to certain treatments. The second was to find new ways of measuring whether or not COPD is getting worse. This would provide new ways of testing whether a new treatment is working.

SPIROMICS I had three sub studies and two key ancillary studies.

Sub studies:

1. Repeatability Substudy: The entire baseline clinic visit was repeated on 100 participants on a volunteer basis. The goal of this substudy was to determine reliability of measurement procedures.
2. Bronchoscopy Substudy: ~300 participants were enrolled for two additional study visits, including a bronchoscopy. The goal of this substudy was to collect and assess biological specimens and relate those results to clinical measurements.
3. Exacerbation Substudy: ~400 participants were enrolled in this substudy. A daily symptom diary was collected on all participants. Participants were also seen in the clinic during a pulmonary exacerbation. The goals of this substudy were to 1) better understand the relationship between symptoms and exacerbations and 2) obtain clinical data and specimens during a pulmonary exacerbation.

Ancillary Studies:

1. Air Pollution Ancillary Study: The SPIROMICS Air Pollution ancillary study used state-of-the art air pollution exposure assessments to determine individual-level outdoor and indoor air pollution exposure. The goals of this substudy were to determine the effect of long-term air pollution exposure on COPD morbidity and to determine whether short-term changes in outdoor air pollution are associated with changes in COPD morbidity.
2. Parametric Response Mapping in COPD: The Parametric Response Mapping (PRM) in COPD ancillary study collected an additional CT scan during the final study visit and used a new analysis technique (PRM) to assess the functional small airways of the lung and emphysema.

Description of SPIROMICS II:

Aim 1 was to define the natural history of "smokers with symptoms despite preserved spirometry" and characterize the airway mucus abnormalities underlying this condition. Aim 2 was to determine the radiographic precursor lesion(s) for emphysema and identify the molecular phenotypes underlying airway disease and emphysema. Aim 3 was to advance understanding of the biology of COPD exacerbations through analysis of predisposing baseline phenotypes, exacerbation triggers and host inflammatory response.

SPIROMICS II continued follow-up of active participants, with no new enrollment. Each participant had one clinic visit at 5-7 years of follow-up from SPIROMICS I baseline and was contacted by telephone every 4 months to assess respiratory health status.

Description of SPIROMICS III:

Aim 1 is to identify the main forms of smoking-related airway disease that are caused by pathological airway mucus, their biological underpinnings, and their physiological significance. Aim 2 is to identify longitudinal trajectories in established and novel CT measures of emphysema, test how they predict COPD progression, and define their underlying biology. Aim 3 is to identify environmental and social determinants of health that impact disease severity and progression and their influence on lung structure, biology, and health disparities in COPD.

SPIROMICS III will enroll and consent approximately 1800 participants to conduct (a) a single in-person clinic visit at approximately 11-16 years of follow-up for those originally enrolled into SPIROMICS I and approximately 5-6 years of follow-up for those originally enrolled into SOURCE (and MAP COPD) (NCT05033990), (b) follow-up telephone calls every 4 months to assess respiratory health status, and (c) to assess indoor and outdoor environmental monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 at baseline visit
* Never smokers: <1 pack-year history of smoking
* Never smokers: Must meet lung function criteria based on spirometry without inhaled bronchodilators
* Current or former smokers: >20 pack-year history of smoking
* Current or former smokers: Must meet lung function criteria based on spirometry with inhaled bronchodilators

Exclusion Criteria:

* Dementia or other cognitive dysfunction which in the opinion of the investigator would prevent the participant from consenting to the study or completing study procedures
* Plans to leave the area in the next 3 years
* Smoking history of > 1 pack-year but <21 pack-years
* BMI > 40 kg/m2 at baseline exam
* Prior significant difficulties with pulmonary function testing
* Hypersensitivity to or intolerance of albuterol sulfate or ipratropium bromide or propellants or excipients of the inhalers
* Non-COPD obstructive lung disease, severe kyphoscoliosis, neuromuscular weakness, or other conditions, including clinically significant cardiovascular and pulmonary disease, that, limit the interpretability of the pulmonary function measures.
* History of Interstitial lung disease
* History of Lung volume reduction surgery or lung resection
* History of lung or other organ transplant
* History of endobronchial valve therapy
* History of large thoracic metal implants (e.g., AICD (automatic implantable cardioverter/defibrillator) and/or pacemaker)
* Currently taking >=10mg a day/20mg every other day of prednisone or equivalent systemic corticosteroid
* Currently taking any immunosuppressive agent
* Current illicit substance abuse, excluding marijuana
* History of or current use of IV Ritalin
* History of or current use of heroin
* History of illegal IV drug use within the last 10 years or more than 5 instances of illegal IV drug use ever
* Known HIV/AIDS infection
* History of lung cancer or any cancer that spread to multiple locations in the body
* History of or current exposure to chemotherapy or radiation treatments that, in the opinion of the investigator, limits the interpretability of the pulmonary function measures.
* Diagnosis of unstable cardiovascular disease including myocardial infarction in the past 6 weeks, uncontrolled congestive heart failure, or uncontrolled arrhythmia
* Any illness expected to cause mortality in the next 3 years
* Active pulmonary infection, including tuberculosis
* History of pulmonary embolism in the past 2 years
* Known diagnosis of primary bronchiectasis
* Currently institutionalized (e.g., prisons, long-term care facilities)
* Known to be a first degree relative of another, already enrolled participant (i.e., biological parent, biological sibling)
* Never smokers only: Current diagnosis of asthma
* Women only: Cannot be pregnant at baseline or plan to become pregnant during the course of the study

Temporal Exclusion Criteria for SPIROMICS III:

* Participants who present with a pulmonary exacerbation, either solely participant-identified or that has been clinically treated, in the last six weeks, can complete the study visit once a six-week window has passed.
* Participants who present with an upper respiratory infection, either solely participant-identified or that has been clinically treated, in the last six weeks, can complete the study visit once a six-week window has passed.
* Participants who present with current use of acute antibiotics or steroids can complete the study visit ≥30 days after discontinuing acute antibiotics/steroids. This does not apply to participants who are on chronic prednisone therapy of <10 mg per day or <20 mg every other day or participants who are currently on chronic, prophylactic, or suppressive antibiotic therapy.
* Participants who present with a myocardial infarction or eye, chest or abdominal surgery within six weeks can complete the study visit after a six-week window has passed.
* Female participants who present <3 months after giving birth will be asked to schedule the visit once three months have passed post-delivery.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Never-smokers, current and former smokers without COPD, and current and former smokers with COPD with access to one of the study clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 2981 (Actual)
Dates: Start 2010-11; Primary Completion 2031-06-17 (Estimated); Study Completion 2031-06-17 (Estimated)

PRIMARY OUTCOMES:
Morbidity | Through study completion, an average of 18 years.
  Morbidity in SPIROMICS will primarily be measured by assessing acute exacerbations in the SPIROMICS cohort.
Lung Function | Through study completion, an average of 18 years.
  COPD is characterized by physiological problems, such as airflow limitations and abnormalities of gas exchange and lung hyperinflation. These features of lung function are accessed objectively in the laboratory setting using spirometry/plethysmography, which can measure such parameters as FEV1 (forced expiratory volume in one second), FVC (forced vital capacity or total volume of air exhaled after full inspiration), FRC (functional residual capacity or volume of gas remaining in the lung at the end of tidal expiration), and IC (inspiratory capacity or maximum volume of gas that can be inspired from end-tidal expiration). The FDA preferred primary endpoint for assessment of alteration in disease progression in COPD is serial measurements of FEV1 over three years.
Mortality | Through study completion, an average of 18 years.
  Deaths of SPIROMICS participants will be identified during follow-up calls and attempts to schedule clinic exams during the three-year study period, and deaths will be recorded in the clinical database. The cause of death will be determined via chart review and adjudication, and deaths attributable to COPD worsening or exacerbation will be recorded as confirmed clinical endpoints, in addition to contributing to the endpoint of all-cause mortality.
SPIROMICS III: Radiology - Emphysema Volume | Through study completion, an average of 18 years.
  Percent Emphysema (percent <-950HU)
SPIROMICS III: Radiology - Functional Small Airway Disease through Parametric Response Mapping (PRM) | Through study completion, an average of 18 years.
  PRM metrics will be used to non-invasively evaluate the regional structural heterogeneity of the lung, including small airways disease and emphysema, and its relationship to clinical measurements. The metric is PRMfSAD.
SPIROMICS III: Radiology - Functional Small Airway Disease through Disease Probability Method (DPM) | Through study completion, an average of 18 years.
  Patients undergo both full-inspiration and full-expiration chest CT scans. These scans are coregistered-aligned voxel-by-voxel-to allow for direct comparison of lung tissue characteristics between breathing phases. Each voxel (3D pixel) in the lung is classified into one of three categories: Normal: No signs of disease, Emphysema: Identified by low attenuation on inspiratory CT, Gas Trapping (SAD): Identified by abnormal retention of air on expiratory CT without emphysema features. The proportion of voxels classified as emphysema, gas trapping, or normal is calculated.
SPIROMICS III: Radiology - Airway Wall Thickness | Through study completion, an average of 18 years.
  Pi10 as a measure of airway wall thickness
SPIROMICS III: Physiology - Lung function (Spirometry) | Through study completion, an average of 18 years.
  Lung function will be assessed as FEV1 through spirometry using forced and slow vital capacity before and after bronchodilator (BD) administration.
SPIROMICS III: Physiology - Lung function (Respiratory Oscillometry) | Through study completion, an average of 18 years.
  Assessment of lung function through respiratory oscillometry.
SPIROMICS III: Biological - Mucin concentrations | Through study completion, an average of 18 years.
  Mucus samples obtained from sputum, bronchial brushings, and Bronchoalveolar Lavage (BAL) will be analyzed for total mucin concentration.
SPIROMICS III: Biological - MUCQ index | Through study completion, an average of 18 years.
  The MUCQ index which integrates mucin concentration with MUC5AC/MUC5B ratios will be calculated and provide more detailed understanding of mucin composition and regulation. The formula MUCQ=[total mucin] x [5AC]/[MUC5B] / 100 will be used.
SPIROMICS III: Biological - Mucin-interacting proteins | Through study completion, an average of 18 years.
  Mucin-interacting proteins will be identified and quantified using labeled and label free mass spectrometry.
SPIROMICS III: Environmental and Social Determinants of Health - Outdoor concentrations of particulate matter (PM) 2.5 | Through study completion, an average of 18 years.
  Data on ambient air quality will be obtained from the EPA DataMart for sites nearest each participant home address. Data will be obtained at the highest temporal resolution and averaged to daily and weekly values. Outdoor concentrations of PM2.5 will be measured in micrograms per cubic meter of air (µg/m³).
SPIROMICS III: Environmental and Social Determinants of Health - Outdoor concentrations of nitrogen dioxide (NO2) | Through study completion, an average of 18 years.
  Data on ambient air quality will be obtained from the EPA DataMart for sites nearest each participant home address. Data will be obtained at the highest temporal resolution and averaged to daily and weekly values. Outdoor concentrations of NO2 will be measured in parts per billion (ppb).
SPIROMICS III: Environmental and Social Determinants of Health - Outdoor concentrations of nitrogen oxides (NOx) | Through study completion, an average of 18 years.
  Data on ambient air quality will be obtained from the EPA DataMart for sites nearest each participant home address. Data will be obtained at the highest temporal resolution and averaged to daily and weekly values. Outdoor concentrations of NOx will be measured in parts per billion (ppb).
SPIROMICS III: Environmental and Social Determinants of Health - Outdoor concentrations of ozone (O3) | Through study completion, an average of 18 years.
  Data on ambient air quality will be obtained from the EPA DataMart for sites nearest each participant home address. Data will be obtained at the highest temporal resolution and averaged to daily and weekly values. Outdoor concentrations of ozone will be measured in parts per billion (ppb).
SPIROMICS III: Environmental and Social Determinants of Health - Outdoor concentrations of wildfire-derived particulate matter (PM) 2.5 | Through study completion, an average of 18 years.
  Data on ambient air quality will be obtained from the EPA DataMart for sites nearest each participant home address. Data will be obtained at the highest temporal resolution and averaged to daily and weekly values. Outdoor concentrations of wildfire-derived PM2.5 will be measured in micrograms per cubic meter of air (µg/m³).
SPIROMICS III: Environmental and Social Determinants of Health - Indoor concentrations of particulate matter (PM) | Through study completion, an average of 18 years.
  Indoor PM will be measured using a low-cost sensor monitor. Monitors will provide a year-long continuous in-home air monitoring and assessment. Indoor concentrations of PM2.5 will be measured in micrograms per cubic meter of air (µg/m³).
SPIROMICS III: Environmental and Social Determinants of Health - Indoor measurements of temperature | Through study completion, an average of 18 years.
  Indoor temperature will be measured using a low-cost sensor monitor. Monitors will provide a year-long continuous in-home air monitoring and assessment.
SPIROMICS III: Environmental and Social Determinants of Health - Indoor measurements of humidity | Through study completion, an average of 18 years.
  Indoor humidity will be measured using a low-cost sensor monitor. Monitors will provide a year-long continuous in-home air monitoring and assessment.
SPIROMICS III: Environmental and Social Determinants of Health - Indoor measurements of NO2 | Through study completion, an average of 18 years.
  Airborne NO2 will be monitored with passive samplers for approximately one week or seven days in the home. Temperature and humidity measurements will be used to adjust the NO2 analytical results as appropriate. Indoor concentrations of NO2 will be measured in parts per billion (ppb).
SPIROMICS III: Environmental and Social Determinants of Health - Indoor measurements of air nicotine | Through study completion, an average of 18 years.
  Air nicotine will be monitored using passive sampling badges for one week or seven days in the home. Nicotine is collected by passive diffusion onto glass fiber filters treated with a 4% sodium bisulfate solution. The cassette is sealed and returned to the clinic laboratory for extraction and analysis. Indoor concentrations of airborne nicotine will be measured in micrograms per cubic meter (µg/m³).
SPIROMICS III: Environmental and Social Determinants of Health - Indoor measurements of settled dust | Through study completion, an average of 18 years.
  Settled dust samples will be collected from the home to ascertain exposure to common household allergens. The presence of indoor allergens will be assessed by extracting protein from the settled dust samples and quantifying them using enzyme-linked immunosorbent assay (ELISA).
SPIROMICS III: Environmental and Social Determinants of Health - Geocoding | Through study completion, an average of 18 years.
  Geocoding will assess residential mobility and neighborhood characteristics including area deprivation, food access, and segregation.
SPIROMICS III: Epigenetic | Through study completion, an average of 18 years.
  Illumina EPIC Methylation Arrays

SECONDARY OUTCOMES:
Repeatability Substudy: Repeatability of clinic visit measurements | Up to end of recruitment (2-6 week measurement repeatability)
  The repeatability of clinic visit measurements will be assessed at the end of this substudy. In this substudy all clinic procedures and samples are repeated/recollected 2-6 weeks after the baseline clinic visit in a subset of participants. This provides a measurement of short-term repeatability of these assessments.
Exacerbation Substudy: Nasal swab analyses | Through study completion, an average of 18 years.
  Self-administered nasal swabs will be collected during an acute exacerbation in a subset of participants. These will be used to better understand the biological processes underlying an acute exacerbation, including providing information about viral triggers and the host inflammatory response. Analyses will include measurements for RNA and DNA.
Exacerbation Substudy: Sputum analyses for ribonucleic acid (RNA) | Through study completion, an average of 18 years.
  Spontaneous sputum will be collected during an acute exacerbation in a subset of participants. It will be used to better understand the biological processes underlying an acute exacerbation, including initial characterization of the host response. Sputum will be analyzed for RNA and host gene expression.
Exacerbation Substudy: Sputum analyses for mucins | Through study completion, an average of 18 years.
  Spontaneous sputum will be collected during an acute exacerbation in a subset of participants. It will be used to better understand the biological processes underlying an acute exacerbation, including initial characterization of the host response. Sputum will be analyzed for mucins.
Exacerbation Substudy: Sputum analyses for proteins | Through study completion, an average of 18 years.
  Spontaneous sputum will be collected during an acute exacerbation in a subset of participants. It will be used to better understand the biological processes underlying an acute exacerbation, including initial characterization of the host response. Sputum will be analyzed for proteins.
Exacerbation Substudy: Sputum analyses for cytokines | Through study completion, an average of 18 years.
  Spontaneous sputum will be collected during an acute exacerbation in a subset of participants. It will be used to better understand the biological processes underlying an acute exacerbation, including initial characterization of the host response. Sputum will be analyzed for cytokines.
Exacerbation Substudy: Assess symptomatic changes in COPD in relation to acute exacerbation | Through study completion, an average of 18 years.
  The exacerbation substudy will collect a daily symptom diary. Data from this daily diary will be used to characterize the stable versus exacerbative state in a subset of participants.

CONTACTS AND LOCATIONS:
Overall Officials: David Couper, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Graham Barr, PhD, MD, Principal Investigator — Columbia University; Robert Paine, MD, Principal Investigator — University of Utah; Eric Hoffman, MD, Principal Investigator — University of Iowa; Prescott Woodruff, MD, Study Chair — University of California at San Francisco; Igor Barjaktarevic, MD, Principal Investigator — University of California at Los Angeles; MeiLan Han, MD, Principal Investigator — University of Michigan; Claudia Onofrei, MD, MSc, Principal Investigator — National Jewish Health; Alejandro Cornellas, MD, Principal Investigator — University of Iowa; Nathaniel Marchetti, DO, Principal Investigator — Temple University; J. Michael Wells, MD, Principal Investigator — University of Alabama at Birmingham; Nadia Hansel, MD, Principal Investigator — Johns Hopkins University; Jerry Krishnan, MD, Principal Investigator — University of Illinois at Chicago; Jessica Bon, MD, MS, ATSF, Principal Investigator — Wake Forest University; Robert Kaner, MD, Principal Investigator — Weill Medical College of Cornell University; Victor Ortega, MD, PhD, Principal Investigator — Mayo Clinic; Christopher Cooper, MD, PhD, Principal Investigator — University of California at Los Angeles; Neil Alexis, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Sanjiv Shah, Principal Investigator — Northwestern University; Joao Lima, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California at Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medicine, New York, New York
  - Columbia University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data and biospecimens collected in SPIROMICS I were submitted to the NHLBI data and biospecimen repository known as BioLINCC. Data, including genetics and genomics, from SPIROMICS I and SPIROMICS II are submitted to the NIH data repository known as dbGaP. All data and biospecimens are also available through the SPIROMICS Genomics and Informatics Center (GIC) at the Collaborative Studies Coordinating Center (CSCC) at The University of North Carolina at Chapel Hill, by request, and according to study policies and procedures.
Supporting Information: Study Protocol
Time Frame: Data and biospecimens from SPIROMICS I and SPIROMICS II are currently available and will remain available indefinitely. The same for data and biospecimens from SPIROMICS III on an annual basis.
Access Criteria: Access criteria for data from BioLINCC are determined by NHLBI, not by the SPIROMICS Investigators.
  Criteria, policies, and procedures for obtaining data and biospecimens directly from the SPIROMICS Genomics and Informatics Center (GIC) at the Collaborative Studies Coordinating Center (CSCC) at The University of North Carolina at Chapel Hill are available on the web site listed below.
URL: https://www.spiromics.org/spiromics/obtaining-data

REFERENCES:
- [Background] Couper D, LaVange LM, Han M, Barr RG, Bleecker E, Hoffman EA, Kanner R, Kleerup E, Martinez FJ, Woodruff PG, Rennard S; SPIROMICS Research Group. Design of the Subpopulations and Intermediate Outcomes in COPD Study (SPIROMICS). Thorax. 2014 May;69(5):491-4. doi: 10.1136/thoraxjnl-2013-203897. Epub 2013 Sep 12. PMID 24029743
- [Background] Freeman CM, Crudgington S, Stolberg VR, Brown JP, Sonstein J, Alexis NE, Doerschuk CM, Basta PV, Carretta EE, Couper DJ, Hastie AT, Kaner RJ, O'Neal WK, Paine R 3rd, Rennard SI, Shimbo D, Woodruff PG, Zeidler M, Curtis JL. Design of a multi-center immunophenotyping analysis of peripheral blood, sputum and bronchoalveolar lavage fluid in the Subpopulations and Intermediate Outcome Measures in COPD Study (SPIROMICS). J Transl Med. 2015 Jan 27;13:19. doi: 10.1186/s12967-014-0374-z. PMID 25622723
- [Background] Sieren JP, Newell JD Jr, Barr RG, Bleecker ER, Burnette N, Carretta EE, Couper D, Goldin J, Guo J, Han MK, Hansel NN, Kanner RE, Kazerooni EA, Martinez FJ, Rennard S, Woodruff PG, Hoffman EA; SPIROMICS Research Group. SPIROMICS Protocol for Multicenter Quantitative Computed Tomography to Phenotype the Lungs. Am J Respir Crit Care Med. 2016 Oct 1;194(7):794-806. doi: 10.1164/rccm.201506-1208PP. PMID 27482984
- [Background] Hansel NN, Paulin LM, Gassett AJ, Peng RD, Alexis N, Fan VS, Bleecker E, Bowler R, Comellas AP, Dransfield M, Han MK, Kim V, Krishnan JA, Pirozzi C, Cooper CB, Martinez F, Woodruff PG, Breysse PJ, Barr RG, Kaufman JD. Design of the Subpopulations and Intermediate Outcome Measures in COPD (SPIROMICS) AIR Study. BMJ Open Respir Res. 2017 May 18;4(1):e000186. doi: 10.1136/bmjresp-2017-000186. eCollection 2017. PMID 28948026
- [Result] O'Neal WK, Anderson W, Basta PV, Carretta EE, Doerschuk CM, Barr RG, Bleecker ER, Christenson SA, Curtis JL, Han MK, Hansel NN, Kanner RE, Kleerup EC, Martinez FJ, Miller BE, Peters SP, Rennard SI, Scholand MB, Tal-Singer R, Woodruff PG, Couper DJ, Davis SM; SPIROMICS Investigators. Comparison of serum, EDTA plasma and P100 plasma for luminex-based biomarker multiplex assays in patients with chronic obstructive pulmonary disease in the SPIROMICS study. J Transl Med. 2014 Jan 8;12:9. doi: 10.1186/1479-5876-12-9. PMID 24397870
- [Result] Smith BM, Hoffman EA, Rabinowitz D, Bleecker E, Christenson S, Couper D, Donohue KM, Han MK, Hansel NN, Kanner RE, Kleerup E, Rennard S, Barr RG. Comparison of spatially matched airways reveals thinner airway walls in COPD. The Multi-Ethnic Study of Atherosclerosis (MESA) COPD Study and the Subpopulations and Intermediate Outcomes in COPD Study (SPIROMICS). Thorax. 2014 Nov;69(11):987-96. doi: 10.1136/thoraxjnl-2014-205160. Epub 2014 Jun 13. PMID 24928812
- [Result] Boes JL, Hoff BA, Bule M, Johnson TD, Rehemtulla A, Chamberlain R, Hoffman EA, Kazerooni EA, Martinez FJ, Han MK, Ross BD, Galban CJ. Parametric response mapping monitors temporal changes on lung CT scans in the subpopulations and intermediate outcome measures in COPD Study (SPIROMICS). Acad Radiol. 2015 Feb;22(2):186-94. doi: 10.1016/j.acra.2014.08.015. Epub 2014 Nov 4. PMID 25442794
- [Result] Putcha N, Puhan MA, Drummond MB, Han MK, Regan EA, Hanania NA, Martinez CH, Foreman M, Bhatt SP, Make B, Ramsdell J, DeMeo DL, Barr RG, Rennard SI, Martinez F, Silverman EK, Crapo J, Wise RA, Hansel NN. A simplified score to quantify comorbidity in COPD. PLoS One. 2014 Dec 16;9(12):e114438. doi: 10.1371/journal.pone.0114438. eCollection 2014. PMID 25514500
- [Result] Paulin LM, Diette GB, Blanc PD, Putcha N, Eisner MD, Kanner RE, Belli AJ, Christenson S, Tashkin DP, Han M, Barr RG, Hansel NN; SPIROMICS Research Group. Occupational exposures are associated with worse morbidity in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2015 Mar 1;191(5):557-65. doi: 10.1164/rccm.201408-1407OC. PMID 25562375
- [Result] Martinez CH, Diaz AA, Parulekar AD, Rennard SI, Kanner RE, Hansel NN, Couper D, Holm KE, Hoth KF, Curtis JL, Martinez FJ, Hanania NA, Regan EA, Paine R 3rd, Cigolle CT, Han MK; COPDGene and SPIROMICS Investigators. Age-Related Differences in Health-Related Quality of Life in COPD: An Analysis of the COPDGene and SPIROMICS Cohorts. Chest. 2016 Apr;149(4):927-35. doi: 10.1016/j.chest.2015.11.025. Epub 2015 Dec 17. PMID 26836895
- [Result] Putcha N, Barr RG, Han MK, Woodruff PG, Bleecker ER, Kanner RE, Martinez FJ, Smith BM, Tashkin DP, Bowler RP, Eisner MD, Rennard SI, Wise RA, Hansel NN; SPIROMICS Investigators. Understanding the impact of second-hand smoke exposure on clinical outcomes in participants with COPD in the SPIROMICS cohort. Thorax. 2016;71:411-420. doi: 10.1136/thoraxjnl-2015-207487. Epub 2016 Mar 9. PMID 26962015
- [Result] Guo J, Wang C, Chan KS, Jin D, Saha PK, Sieren JP, Barr RG, Han MK, Kazerooni E, Cooper CB, Couper D, Newell JD Jr, Hoffman EA; SPIROMICS Research Group. A controlled statistical study to assess measurement variability as a function of test object position and configuration for automated surveillance in a multicenter longitudinal COPD study (SPIROMICS). Med Phys. 2016 May;43(5):2598. doi: 10.1118/1.4947303. PMID 27147369
- [Result] Woodruff PG, Barr RG, Bleecker E, Christenson SA, Couper D, Curtis JL, Gouskova NA, Hansel NN, Hoffman EA, Kanner RE, Kleerup E, Lazarus SC, Martinez FJ, Paine R 3rd, Rennard S, Tashkin DP, Han MK; SPIROMICS Research Group. Clinical Significance of Symptoms in Smokers with Preserved Pulmonary Function. N Engl J Med. 2016 May 12;374(19):1811-21. doi: 10.1056/NEJMoa1505971. PMID 27168432
- [Result] Sun W, Kechris K, Jacobson S, Drummond MB, Hawkins GA, Yang J, Chen TH, Quibrera PM, Anderson W, Barr RG, Basta PV, Bleecker ER, Beaty T, Casaburi R, Castaldi P, Cho MH, Comellas A, Crapo JD, Criner G, Demeo D, Christenson SA, Couper DJ, Curtis JL, Doerschuk CM, Freeman CM, Gouskova NA, Han MK, Hanania NA, Hansel NN, Hersh CP, Hoffman EA, Kaner RJ, Kanner RE, Kleerup EC, Lutz S, Martinez FJ, Meyers DA, Peters SP, Regan EA, Rennard SI, Scholand MB, Silverman EK, Woodruff PG, O'Neal WK, Bowler RP; SPIROMICS Research Group; COPDGene Investigators. Common Genetic Polymorphisms Influence Blood Biomarker Measurements in COPD. PLoS Genet. 2016 Aug 17;12(8):e1006011. doi: 10.1371/journal.pgen.1006011. eCollection 2016 Aug. PMID 27532455
- [Result] Martinez CH, Diaz AA, Meldrum C, Curtis JL, Cooper CB, Pirozzi C, Kanner RE, Paine R 3rd, Woodruff PG, Bleecker ER, Hansel NN, Barr RG, Marchetti N, Criner GJ, Kazerooni EA, Hoffman EA, Ross BD, Galban CJ, Cigolle CT, Martinez FJ, Han MK; SPIROMICS Investigators. Age and Small Airway Imaging Abnormalities in Subjects with and without Airflow Obstruction in SPIROMICS. Am J Respir Crit Care Med. 2017 Feb 15;195(4):464-472. doi: 10.1164/rccm.201604-0871OC. PMID 27564413
- [Result] Keene JD, Jacobson S, Kechris K, Kinney GL, Foreman MG, Doerschuk CM, Make BJ, Curtis JL, Rennard SI, Barr RG, Bleecker ER, Kanner RE, Kleerup EC, Hansel NN, Woodruff PG, Han MK, Paine R 3rd, Martinez FJ, Bowler RP, O'Neal WK; COPDGene and SPIROMICS Investigators double dagger. Biomarkers Predictive of Exacerbations in the SPIROMICS and COPDGene Cohorts. Am J Respir Crit Care Med. 2017 Feb 15;195(4):473-481. doi: 10.1164/rccm.201607-1330OC. PMID 27579823
- [Result] Hobbs BD, de Jong K, Lamontagne M, Bosse Y, Shrine N, Artigas MS, Wain LV, Hall IP, Jackson VE, Wyss AB, London SJ, North KE, Franceschini N, Strachan DP, Beaty TH, Hokanson JE, Crapo JD, Castaldi PJ, Chase RP, Bartz TM, Heckbert SR, Psaty BM, Gharib SA, Zanen P, Lammers JW, Oudkerk M, Groen HJ, Locantore N, Tal-Singer R, Rennard SI, Vestbo J, Timens W, Pare PD, Latourelle JC, Dupuis J, O'Connor GT, Wilk JB, Kim WJ, Lee MK, Oh YM, Vonk JM, de Koning HJ, Leng S, Belinsky SA, Tesfaigzi Y, Manichaikul A, Wang XQ, Rich SS, Barr RG, Sparrow D, Litonjua AA, Bakke P, Gulsvik A, Lahousse L, Brusselle GG, Stricker BH, Uitterlinden AG, Ampleford EJ, Bleecker ER, Woodruff PG, Meyers DA, Qiao D, Lomas DA, Yim JJ, Kim DK, Hawrylkiewicz I, Sliwinski P, Hardin M, Fingerlin TE, Schwartz DA, Postma DS, MacNee W, Tobin MD, Silverman EK, Boezen HM, Cho MH; COPDGene Investigators; ECLIPSE Investigators; LifeLines Investigators; SPIROMICS Research Group; International COPD Genetics Network Investigators; UK BiLEVE Investigators; International COPD Genetics Consortium. Genetic loci associated with chronic obstructive pulmonary disease overlap with loci for lung function and pulmonary fibrosis. Nat Genet. 2017 Mar;49(3):426-432. doi: 10.1038/ng.3752. Epub 2017 Feb 6. PMID 28166215
- [Result] Han MK, Quibrera PM, Carretta EE, Barr RG, Bleecker ER, Bowler RP, Cooper CB, Comellas A, Couper DJ, Curtis JL, Criner G, Dransfield MT, Hansel NN, Hoffman EA, Kanner RE, Krishnan JA, Martinez CH, Pirozzi CB, O'Neal WK, Rennard S, Tashkin DP, Wedzicha JA, Woodruff P, Paine R 3rd, Martinez FJ; SPIROMICS investigators. Frequency of exacerbations in patients with chronic obstructive pulmonary disease: an analysis of the SPIROMICS cohort. Lancet Respir Med. 2017 Aug;5(8):619-626. doi: 10.1016/S2213-2600(17)30207-2. Epub 2017 Jun 28. PMID 28668356
- [Result] Kesimer M, Ford AA, Ceppe A, Radicioni G, Cao R, Davis CW, Doerschuk CM, Alexis NE, Anderson WH, Henderson AG, Barr RG, Bleecker ER, Christenson SA, Cooper CB, Han MK, Hansel NN, Hastie AT, Hoffman EA, Kanner RE, Martinez F, Paine R 3rd, Woodruff PG, O'Neal WK, Boucher RC. Airway Mucin Concentration as a Marker of Chronic Bronchitis. N Engl J Med. 2017 Sep 7;377(10):911-922. doi: 10.1056/NEJMoa1701632. PMID 28877023
- [Result] Bowler RP, Hansel NN, Jacobson S, Graham Barr R, Make BJ, Han MK, O'Neal WK, Oelsner EC, Casaburi R, Barjaktarevic I, Cooper C, Foreman M, Wise RA, DeMeo DL, Silverman EK, Bailey W, Harrington KF, Woodruff PG, Drummond MB; for COPDGene and SPIROMICS Investigators. Electronic Cigarette Use in US Adults at Risk for or with COPD: Analysis from Two Observational Cohorts. J Gen Intern Med. 2017 Dec;32(12):1315-1322. doi: 10.1007/s11606-017-4150-7. Epub 2017 Sep 7. PMID 28884423
- [Result] Martinez CH, Li SX, Hirzel AJ, Stolberg VR, Alexis NE, Barr RG, Bleecker ER, Carretta EE, Christenson SA, Cooper CB, Couper DJ, Doerschuk CM, Han MK, Hansel NN, Hastie AT, Hoffman EA, Kaner RJ, Martinez FJ, Meyers DA, O'Neal WK, Paine R 3rd, Putcha N, Rennard SI, Woodruff PG, Zeidler M, Curtis JL, Freeman CM; SPIROMICS Investigators. Alveolar eosinophilia in current smokers with chronic obstructive pulmonary disease in the SPIROMICS cohort. J Allergy Clin Immunol. 2018 Jan;141(1):429-432. doi: 10.1016/j.jaci.2017.07.039. Epub 2017 Sep 12. PMID 28916185
- [Result] Anderson WH, Ha JW, Couper DJ, O'Neal WK, Barr RG, Bleecker ER, Carretta EE, Cooper CB, Doerschuk CM, Drummond MB, Han MK, Hansel NN, Kim V, Kleerup EC, Martinez FJ, Rennard SI, Tashkin D, Woodruff PG, Paine R 3rd, Curtis JL, Kanner RE; SPIROMICS Research Group. Variability in objective and subjective measures affects baseline values in studies of patients with COPD. PLoS One. 2017 Sep 21;12(9):e0184606. doi: 10.1371/journal.pone.0184606. eCollection 2017. PMID 28934249
- [Result] Bradford E, Jacobson S, Varasteh J, Comellas AP, Woodruff P, O'Neal W, DeMeo DL, Li X, Kim V, Cho M, Castaldi PJ, Hersh C, Silverman EK, Crapo JD, Kechris K, Bowler RP. The value of blood cytokines and chemokines in assessing COPD. Respir Res. 2017 Oct 24;18(1):180. doi: 10.1186/s12931-017-0662-2. PMID 29065892
- [Result] Hastie AT, Martinez FJ, Curtis JL, Doerschuk CM, Hansel NN, Christenson S, Putcha N, Ortega VE, Li X, Barr RG, Carretta EE, Couper DJ, Cooper CB, Hoffman EA, Kanner RE, Kleerup E, O'Neal WK, Paine R 3rd, Peters SP, Alexis NE, Woodruff PG, Han MK, Meyers DA, Bleecker ER; SPIROMICS investigators. Association of sputum and blood eosinophil concentrations with clinical measures of COPD severity: an analysis of the SPIROMICS cohort. Lancet Respir Med. 2017 Dec;5(12):956-967. doi: 10.1016/S2213-2600(17)30432-0. Epub 2017 Nov 13. PMID 29146301
- [Result] Smith BM, Traboulsi H, Austin JHM, Manichaikul A, Hoffman EA, Bleecker ER, Cardoso WV, Cooper C, Couper DJ, Dashnaw SM, Guo J, Han MK, Hansel NN, Hughes EW, Jacobs DR Jr, Kanner RE, Kaufman JD, Kleerup E, Lin CL, Liu K, Lo Cascio CM, Martinez FJ, Nguyen JN, Prince MR, Rennard S, Rich SS, Simon L, Sun Y, Watson KE, Woodruff PG, Baglole CJ, Barr RG; MESA Lung and SPIROMICS investigators. Human airway branch variation and chronic obstructive pulmonary disease. Proc Natl Acad Sci U S A. 2018 Jan 30;115(5):E974-E981. doi: 10.1073/pnas.1715564115. Epub 2018 Jan 16. PMID 29339516
- [Result] Fawzy A, Putcha N, Paulin LM, Aaron CP, Labaki WW, Han MK, Wise RA, Kanner RE, Bowler RP, Barr RG, Hansel NN; SPIROMICS and COPDGene Investigators. Association of thrombocytosis with COPD morbidity: the SPIROMICS and COPDGene cohorts. Respir Res. 2018 Jan 26;19(1):20. doi: 10.1186/s12931-018-0717-z. PMID 29373977
- [Result] Fernandez-Baldera A, Hatt CR, Murray S, Hoffman EA, Kazerooni EA, Martinez FJ, Han MK, Galban CJ. Correcting Nonpathological Variation in Longitudinal Parametric Response Maps of CT Scans in COPD Subjects: SPIROMICS. Tomography. 2017 Sep;3(3):138-145. doi: 10.18383/j.tom.2017.00013. PMID 29457137
- [Result] Han MK, Tayob N, Murray S, Woodruff PG, Curtis JL, Kim V, Criner G, Galban CJ, Ross BD, Hoffman EA, Lynch DA, Kazerooni E, Martinez FJ; COPDGene and SPIROMICS Investigators. Association between Emphysema and Chronic Obstructive Pulmonary Disease Outcomes in the COPDGene and SPIROMICS Cohorts: A Post Hoc Analysis of Two Clinical Trials. Am J Respir Crit Care Med. 2018 Jul 15;198(2):265-267. doi: 10.1164/rccm.201801-0051LE. No abstract available. PMID 29485901
- [Result] Zeidler MR, Martin JL, Kleerup EC, Schneider H, Mitchell MN, Hansel NN, Sundar K, Schotland H, Basner RC, Wells JM, Krishnan JA, Criner GJ, Cristenson S, Krachman S, Badr MS; SPIROMICS Research Group. Sleep disruption as a predictor of quality of life among patients in the subpopulations and intermediate outcome measures in COPD study (SPIROMICS). Sleep. 2018 May 1;41(5):zsy044. doi: 10.1093/sleep/zsy044. PMID 29534240
- [Result] Burkes RM, Gassett AJ, Ceppe AS, Anderson W, O'Neal WK, Woodruff PG, Krishnan JA, Barr RG, Han MK, Martinez FJ, Comellas AP, Lambert AA, Kaufman JD, Dransfield MT, Wells JM, Kanner RE, Paine R 3rd, Bleecker ER, Paulin LM, Hansel NN, Drummond MB; Current and former investigators of the SPIROMICS sites and reading centers. Rural Residence and Chronic Obstructive Pulmonary Disease Exacerbations. Analysis of the SPIROMICS Cohort. Ann Am Thorac Soc. 2018 Jul;15(7):808-816. doi: 10.1513/AnnalsATS.201710-837OC. PMID 29584453
- [Result] Morris MA, Jacobson SR, Kinney GL, Tashkin DP, Woodruff PG, Hoffman EA, Kanner RE, Cooper CB, Drummond MB, Barr RG, Oelsner EC, Make BJ, Han MK, Hansel NN, O'Neal WK, Bowler RP. Marijuana Use Associations with Pulmonary Symptoms and Function in Tobacco Smokers Enrolled in the Subpopulations and Intermediate Outcome Measures in COPD Study (SPIROMICS). Chronic Obstr Pulm Dis. 2018 Jan 24;5(1):46-56. doi: 10.15326/jcopdf.5.1.2017.0141. PMID 29629404
- [Result] Putcha N, Paul GG, Azar A, Wise RA, O'Neal WK, Dransfield MT, Woodruff PG, Curtis JL, Comellas AP, Drummond MB, Lambert AA, Paulin LM, Fawzy A, Kanner RE, Paine R 3rd, Han MK, Martinez FJ, Bowler RP, Barr RG, Hansel NN; SPIROMICS investigators. Lower serum IgA is associated with COPD exacerbation risk in SPIROMICS. PLoS One. 2018 Apr 12;13(4):e0194924. doi: 10.1371/journal.pone.0194924. eCollection 2018. PMID 29649230
- [Result] Labaki WW, Xia M, Murray S, Curtis JL, Barr RG, Bhatt SP, Bleecker ER, Hansel NN, Cooper CB, Dransfield MT, Wells JM, Hoffman EA, Kanner RE, Paine R 3rd, Ortega VE, Peters SP, Krishnan JA, Bowler RP, Couper DJ, Woodruff PG, Martinez FJ, Martinez CH, Han MK. NT-proBNP in stable COPD and future exacerbation risk: Analysis of the SPIROMICS cohort. Respir Med. 2018 Jul;140:87-93. doi: 10.1016/j.rmed.2018.06.005. Epub 2018 Jun 5. PMID 29957287
- [Result] Li X, Ortega VE, Ampleford EJ, Graham Barr R, Christenson SA, Cooper CB, Couper D, Dransfield MT, Han MLK, Hansel NN, Hoffman EA, Kanner RE, Kleerup EC, Martinez FJ, Paine R 3rd, Woodruff PG, Hawkins GA, Bleecker ER, Meyers DA; SPIROMICS Research Group. Genome-wide association study of lung function and clinical implication in heavy smokers. BMC Med Genet. 2018 Aug 1;19(1):134. doi: 10.1186/s12881-018-0656-z. PMID 30068317
- [Result] Kesimer M, Smith BM, Ceppe A, Ford AA, Anderson WH, Barr RG, O'Neal WK, Boucher RC; SPIROMICS Investigative Group. Mucin Concentrations and Peripheral Airway Obstruction in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2018 Dec 1;198(11):1453-1456. doi: 10.1164/rccm.201806-1016LE. No abstract available. PMID 30130124
- [Result] Ghosh S, Anderson WH, Putcha N, Han MK, Curtis JL, Criner GJ, Dransfield MT, Barr RG, Krishnan JA, Lazarus SC, Cooper CB, Paine R 3rd, Peters SP, Hansel NN, Martinez FJ, Drummond MB; Current and former investigators of the SPIROMICS sites and reading centers. Alignment of Inhaled Chronic Obstructive Pulmonary Disease Therapies with Published Strategies. Analysis of the Global Initiative for Chronic Obstructive Lung Disease Recommendations in SPIROMICS. Ann Am Thorac Soc. 2019 Feb;16(2):200-208. doi: 10.1513/AnnalsATS.201804-283OC. PMID 30216731
- [Result] Haghighi B, Choi S, Choi J, Hoffman EA, Comellas AP, Newell JD Jr, Graham Barr R, Bleecker E, Cooper CB, Couper D, Han ML, Hansel NN, Kanner RE, Kazerooni EA, Kleerup EAC, Martinez FJ, O'Neal W, Rennard SI, Woodruff PG, Lin CL. Imaging-based clusters in current smokers of the COPD cohort associate with clinical characteristics: the SubPopulations and Intermediate Outcome Measures in COPD Study (SPIROMICS). Respir Res. 2018 Sep 18;19(1):178. doi: 10.1186/s12931-018-0888-7. PMID 30227877
- [Result] Paulin LM, Smith BM, Koch A, Han M, Hoffman EA, Martinez C, Ejike C, Blanc PD, Rous J, Barr RG, Peters SP, Paine R 3rd, Pirozzi C, Cooper CB, Dransfield MT, Comellas AP, Kanner RE, Drummond MB, Putcha N, Hansel NN. Occupational Exposures and Computed Tomographic Imaging Characteristics in the SPIROMICS Cohort. Ann Am Thorac Soc. 2018 Dec;15(12):1411-1419. doi: 10.1513/AnnalsATS.201802-150OC. PMID 30339479
- [Result] Christenson SA, van den Berge M, Faiz A, Inkamp K, Bhakta N, Bonser LR, Zlock LT, Barjaktarevic IZ, Barr RG, Bleecker ER, Boucher RC, Bowler RP, Comellas AP, Curtis JL, Han MK, Hansel NN, Hiemstra PS, Kaner RJ, Krishnanm JA, Martinez FJ, O'Neal WK, Paine R 3rd, Timens W, Wells JM, Spira A, Erle DJ, Woodruff PG. An airway epithelial IL-17A response signature identifies a steroid-unresponsive COPD patient subgroup. J Clin Invest. 2019 Jan 2;129(1):169-181. doi: 10.1172/JCI121087. Epub 2018 Nov 26. PMID 30383540
- [Result] Wells JM, Parker MM, Oster RA, Bowler RP, Dransfield MT, Bhatt SP, Cho MH, Kim V, Curtis JL, Martinez FJ, Paine R 3rd, O'Neal W, Labaki WW, Kaner RJ, Barjaktarevic I, Han MK, Silverman EK, Crapo JD, Barr RG, Woodruff P, Castaldi PJ, Gaggar A; SPIROMICS and COPDGene Investigators. Elevated circulating MMP-9 is linked to increased COPD exacerbation risk in SPIROMICS and COPDGene. JCI Insight. 2018 Nov 15;3(22):e123614. doi: 10.1172/jci.insight.123614. PMID 30429371
- [Result] Pirozzi CS, Gu T, Quibrera PM, Carretta EE, Han MK, Murray S, Cooper CB, Tashkin DP, Kleerup EC, Barjaktarevic I, Hoffman EA, Martinez CH, Christenson SA, Hansel NN, Graham Barr R, Bleecker ER, Ortega VE, Martinez FJ, Kanner RE, Paine R 3rd; NHLBI SubPopulations and InteRmediate Outcome Measures In COPD Study (SPIROMICS). Heterogeneous burden of lung disease in smokers with borderline airflow obstruction. Respir Res. 2018 Nov 20;19(1):223. doi: 10.1186/s12931-018-0911-z. PMID 30454050
- [Result] Bhatt SP, Nath HP, Kim YI, Ramachandran R, Watts JR, Terry NLJ, Sonavane S, Deshmane SP, Woodruff PG, Oelsner EC, Bodduluri S, Han MK, Labaki WW, Michael Wells J, Martinez FJ, Barr RG, Dransfield MT; SPIROMICS investigators. Centrilobular emphysema and coronary artery calcification: mediation analysis in the SPIROMICS cohort. Respir Res. 2018 Dec 18;19(1):257. doi: 10.1186/s12931-018-0946-1. PMID 30563576
- [Result] Fawzy A, Putcha N, Aaron CP, Bowler RP, Comellas AP, Cooper CB, Dransfield MT, Han MK, Hoffman EA, Kanner RE, Krishnan JA, Labaki WW, Paine R 3rd, Paulin LM, Peters SP, Wise R, Barr RG, Hansel NN; SPIROMICS Investigators. Aspirin Use and Respiratory Morbidity in COPD: A Propensity Score-Matched Analysis in Subpopulations and Intermediate Outcome Measures in COPD Study. Chest. 2019 Mar;155(3):519-527. doi: 10.1016/j.chest.2018.11.028. Epub 2018 Dec 26. PMID 30593776
- [Result] Wells JM, Arenberg DA, Barjaktarevic I, Bhatt SP, Bowler RP, Christenson SA, Couper DJ, Dransfield MT, Han MK, Hoffman EA, Kaner RJ, Kim V, Kleerup E, Martinez FJ, Moore WC, O'Beirne SL, Paine R 3rd, Putcha N, Raman SM, Barr RG, Rennard SI, Woodruff PG, Curtis JL. Safety and Tolerability of Comprehensive Research Bronchoscopy in Chronic Obstructive Pulmonary Disease. Results from the SPIROMICS Bronchoscopy Substudy. Ann Am Thorac Soc. 2019 Apr;16(4):439-446. doi: 10.1513/AnnalsATS.201807-441OC. PMID 30653926
- [Result] Garudadri S, Woodruff PG, Han MK, Curtis JL, Barr RG, Bleecker ER, Bowler RP, Comellas A, Cooper CB, Criner G, Dransfield MT, Hansel NN, Paine R 3rd, Krishnan JA, Peters SP, Hastie AT, Martinez FJ, O'Neal WK, Couper DJ, Alexis NE, Christenson SA. Systemic Markers of Inflammation in Smokers With Symptoms Despite Preserved Spirometry in SPIROMICS. Chest. 2019 May;155(5):908-917. doi: 10.1016/j.chest.2018.12.022. Epub 2019 Jan 23. PMID 30684474
- [Result] Putcha N, Fawzy A, Paul GG, Lambert AA, Psoter KJ, Sidhaye VK, Woo J, Wells JM, Labaki WW, Doerschuk CM, Kanner RE, Han MK, Martinez C, Paulin LM, Martinez FJ, Wise RA, O'Neal WK, Barr RG, Hansel NN; SPIROMICS investigators. Anemia and Adverse Outcomes in a Chronic Obstructive Pulmonary Disease Population with a High Burden of Comorbidities. An Analysis from SPIROMICS. Ann Am Thorac Soc. 2018 Jun;15(6):710-717. doi: 10.1513/AnnalsATS.201708-687OC. PMID 30726108
- [Result] Oelsner EC, Ortega VE, Smith BM, Nguyen JN, Manichaikul AW, Hoffman EA, Guo X, Taylor KD, Woodruff PG, Couper DJ, Hansel NN, Martinez FJ, Paine R 3rd, Han MK, Cooper C, Dransfield MT, Criner G, Krishnan JA, Bowler R, Bleecker ER, Peters S, Rich SS, Meyers DA, Rotter JI, Barr RG. A Genetic Risk Score Associated with Chronic Obstructive Pulmonary Disease Susceptibility and Lung Structure on Computed Tomography. Am J Respir Crit Care Med. 2019 Sep 15;200(6):721-731. doi: 10.1164/rccm.201812-2355OC. PMID 30925230
- [Result] Cho HB, Chae KJ, Jin GY, Choi J, Lin CL, Hoffman EA, Wenzel SE, Castro M, Fain SB, Jarjour NN, Schiebler ML, Barr RG, Hansel N, Cooper CB, Kleerup EC, Han MK, Woodruff PG, Kanner RE, Bleecker ER, Peters SP, Moore WC, Lee CH, Choi S; National Heart, Lung and Blood Institute's SubPopulations and InteRmediate Outcome Measures In COPD Study (SPIROMICS) and Severe Asthma Research Program (SARP). Structural and Functional Features on Quantitative Chest Computed Tomography in the Korean Asian versus the White American Healthy Non-Smokers. Korean J Radiol. 2019 Jul;20(7):1236-1245. doi: 10.3348/kjr.2019.0083. PMID 31270987
- [Result] Haghighi B, Choi S, Choi J, Hoffman EA, Comellas AP, Newell JD Jr, Lee CH, Barr RG, Bleecker E, Cooper CB, Couper D, Han ML, Hansel NN, Kanner RE, Kazerooni EA, Kleerup EAC, Martinez FJ, O'Neal W, Paine R 3rd, Rennard SI, Smith BM, Woodruff PG, Lin CL. Imaging-based clusters in former smokers of the COPD cohort associate with clinical characteristics: the SubPopulations and intermediate outcome measures in COPD study (SPIROMICS). Respir Res. 2019 Jul 15;20(1):153. doi: 10.1186/s12931-019-1121-z. PMID 31307479
- [Result] Halper-Stromberg E, Gillenwater L, Cruickshank-Quinn C, O'Neal WK, Reisdorph N, Petrache I, Zhuang Y, Labaki WW, Curtis JL, Wells J, Rennard S, Pratte KA, Woodruff P, Stringer KA, Kechris K, Bowler RP. Bronchoalveolar Lavage Fluid from COPD Patients Reveals More Compounds Associated with Disease than Matched Plasma. Metabolites. 2019 Jul 25;9(8):157. doi: 10.3390/metabo9080157. PMID 31349744
- [Result] Labaki WW, Gu T, Murray S, Curtis JL, Yeomans L, Bowler RP, Barr RG, Comellas AP, Hansel NN, Cooper CB, Barjaktarevic I, Kanner RE, Paine R 3rd, McDonald MN, Krishnan JA, Peters SP, Woodruff PG, O'Neal WK, Diao W, He B, Martinez FJ, Standiford TJ, Stringer KA, Han MK. Serum amino acid concentrations and clinical outcomes in smokers: SPIROMICS metabolomics study. Sci Rep. 2019 Aug 6;9(1):11367. doi: 10.1038/s41598-019-47761-w. PMID 31388056
- [Result] Arjomandi M, Zeng S, Barjaktarevic I, Barr RG, Bleecker ER, Bowler RP, Buhr RG, Criner GJ, Comellas AP, Cooper CB, Couper DJ, Curtis JL, Dransfield MT, Han MK, Hansel NN, Hoffman EA, Kaner RJ, Kanner RE, Krishnan JA, Paine R 3rd, Peters SP, Rennard SI, Woodruff PG; SPIROMICS Investigators. Radiographic lung volumes predict progression to COPD in smokers with preserved spirometry in SPIROMICS. Eur Respir J. 2019 Oct 31;54(4):1802214. doi: 10.1183/13993003.02214-2018. Print 2019 Oct. PMID 31439683
- [Result] Ortega VE, Li X, O'Neal WK, Lackey L, Ampleford E, Hawkins GA, Grayeski PJ, Laederach A, Barjaktarevic I, Barr RG, Cooper C, Couper D, Han MK, Kanner RE, Kleerup EC, Martinez FJ, Paine R 3rd, Peters SP, Pirozzi C, Rennard SI, Woodruff PG, Hoffman EA, Meyers DA, Bleecker ER; NHLBI Subpopulations and Intermediate Outcomes Measures in COPD Study (SPIROMICS). The Effects of Rare SERPINA1 Variants on Lung Function and Emphysema in SPIROMICS. Am J Respir Crit Care Med. 2020 Mar 1;201(5):540-554. doi: 10.1164/rccm.201904-0769OC. PMID 31661293
- [Result] Wells JM, Xing D, Viera L, Burkes RM, Wu Y, Bhatt SP, Dransfield MT, Couper DJ, O'Neal W, Hoffman EA, Gaggar A, Barjaktarevic I, Curtis JL, Labaki WW, Han MLK, Freeman CM, Putcha N, Schlange T, Blalock JE; SPIROMICS Investigators,. The matrikine acetyl-proline-glycine-proline and clinical features of COPD: findings from SPIROMICS. Respir Res. 2019 Nov 12;20(1):254. doi: 10.1186/s12931-019-1230-8. PMID 31718676
- [Result] Paulin LM, Gassett AJ, Alexis NE, Kirwa K, Kanner RE, Peters S, Krishnan JA, Paine R 3rd, Dransfield M, Woodruff PG, Cooper CB, Barr RG, Comellas AP, Pirozzi CS, Han M, Hoffman EA, Martinez FJ, Woo H, Peng RD, Fawzy A, Putcha N, Breysse PN, Kaufman JD, Hansel NN; for SPIROMICS investigators. Association of Long-term Ambient Ozone Exposure With Respiratory Morbidity in Smokers. JAMA Intern Med. 2020 Jan 1;180(1):106-115. doi: 10.1001/jamainternmed.2019.5498. PMID 31816012
- [Result] Zhang WZ, Rice MC, Hoffman KL, Oromendia C, Barjaktarevic IZ, Wells JM, Hastie AT, Labaki WW, Cooper CB, Comellas AP, Criner GJ, Krishnan JA, Paine R 3rd, Hansel NN, Bowler RP, Barr RG, Peters SP, Woodruff PG, Curtis JL, Han MK, Ballman KV, Martinez FJ, Choi AM, Nakahira K, Cloonan SM, Choi ME; SPIROMICS Investigators. Association of urine mitochondrial DNA with clinical measures of COPD in the SPIROMICS cohort. JCI Insight. 2020 Feb 13;5(3):e133984. doi: 10.1172/jci.insight.133984. PMID 31895696
- [Result] Barjaktarevic IZ, Buhr RG, Wang X, Hu S, Couper D, Anderson W, Kanner RE, Paine Iii R, Bhatt SP, Bhakta NR, Arjomandi M, Kaner RJ, Pirozzi CS, Curtis JL, O'Neal WK, Woodruff PG, Han MK, Martinez FJ, Hansel N, Wells JM, Ortega VE, Hoffman EA, Doerschuk CM, Kim V, Dransfield MT, Drummond MB, Bowler R, Criner G, Christenson SA, Ronish B, Peters SP, Krishnan JA, Tashkin DP, Cooper CB; NHLBI SubPopulations and InteRmediate Outcome Measures In COPD Study (SPIROMICS). Clinical Significance of Bronchodilator Responsiveness Evaluated by Forced Vital Capacity in COPD: SPIROMICS Cohort Analysis. Int J Chron Obstruct Pulmon Dis. 2019 Dec 20;14:2927-2938. doi: 10.2147/COPD.S220164. eCollection 2019. PMID 31908441
- [Result] Burkes RM, Ceppe AS, Doerschuk CM, Couper D, Hoffman EA, Comellas AP, Barr RG, Krishnan JA, Cooper C, Labaki WW, Ortega VE, Wells JM, Criner GJ, Woodruff PG, Bowler RP, Pirozzi CS, Hansel NN, Wise RA, Brown TT, Drummond MB; SPIROMICS Investigators. Associations Among 25-Hydroxyvitamin D Levels, Lung Function, and Exacerbation Outcomes in COPD: An Analysis of the SPIROMICS Cohort. Chest. 2020 Apr;157(4):856-865. doi: 10.1016/j.chest.2019.11.047. Epub 2020 Jan 17. PMID 31958447
- [Result] Stott-Miller M, Mullerova H, Miller B, Tabberer M, El Baou C, Keeley T, Martinez FJ, Han M, Dransfield M, Hansel NN, Cooper CB, Woodruff P, Ortega VE, Comellas AP, Paine Iii R, Kanner RE, Anderson W, Drummond MB, Kim V, Tal-Singer R, Lazaar AL. Defining Chronic Mucus Hypersecretion Using the CAT in the SPIROMICS Cohort. Int J Chron Obstruct Pulmon Dis. 2020 Oct 13;15:2467-2476. doi: 10.2147/COPD.S267002. eCollection 2020. PMID 33116463
- [Result] Burkes RM, Ceppe AS, Couper DJ, Comellas AP, Wells JM, Peters SP, Criner GJ, Kanner RE, Paine R 3rd, Christenson SA, Cooper CB, Barjaktarevic IZ, Krishnan JA, Labaki WW, Han MK, Curtis JL, Hansel NN, Wise RA, Drummond MB; SPIROMICS collaborators. Plasma Cathelicidin is Independently Associated with Reduced Lung Function in COPD: Analysis of the Subpopulations and Intermediate Outcome Measures in COPD Study Cohort. Chronic Obstr Pulm Dis. 2020 Oct;7(4):370-381. doi: 10.15326/jcopdf.7.4.2020.0142. PMID 33108110
- [Result] Ejike CO, Woo H, Galiatsatos P, Paulin LM, Krishnan JA, Cooper CB, Couper DJ, Kanner RE, Bowler RP, Hoffman EA, Comellas AP, Criner GJ, Barr RG, Martinez FJ, Han MK, Martinez CH, Ortega VE, Parekh TM, Christenson SA, Thakur N, Baugh A, Belz DC, Raju S, Gassett AJ, Kaufman JD, Putcha N, Hansel NN. Contribution of Individual and Neighborhood Factors to Racial Disparities in Respiratory Outcomes. Am J Respir Crit Care Med. 2021 Apr 15;203(8):987-997. doi: 10.1164/rccm.202002-0253OC. PMID 33007162
- [Result] Cooper CB, Paine R, Curtis JL, Kanner RE, Martinez CH, Meldrum CA, Bowler R, O'Neal W, Hoffman EA, Couper D, Quibrera M, Criner G, Dransfield MT, Han MK, Hansel NN, Krishnan JA, Lazarus SC, Peters SP, Barr RG, Martinez FJ, Woodruff PG; SPIROMICS investigators. Novel Respiratory Disability Score Predicts COPD Exacerbations and Mortality in the SPIROMICS Cohort. Int J Chron Obstruct Pulmon Dis. 2020 Aug 4;15:1887-1898. doi: 10.2147/COPD.S250191. eCollection 2020. PMID 32821092
- [Result] Zhang WZ, Oromendia C, Kikkers SA, Butler JJ, O'Beirne S, Kim K, O'Neal WK, Freeman CM, Christenson SA, Peters SP, Wells JM, Doerschuk C, Putcha N, Barjaktarevic I, Woodruff PG, Cooper CB, Bowler RP, Comellas AP, Criner GJ, Paine R 3rd, Hansel NN, Han MK, Crystal RG, Kaner RJ, Ballman KV, Curtis JL, Martinez FJ, Cloonan SM. Increased airway iron parameters and risk for exacerbation in COPD: an analysis from SPIROMICS. Sci Rep. 2020 Jun 29;10(1):10562. doi: 10.1038/s41598-020-67047-w. PMID 32601308
- [Result] Galiatsatos P, Woo H, Paulin LM, Kind A, Putcha N, Gassett AJ, Cooper CB, Dransfield MT, Parekh TM, Oates GR, Barr RG, Comellas AP, Han MK, Peters SP, Krishnan JA, Labaki WW, McCormack MC, Kaufman JD, Hansel NN. The Association Between Neighborhood Socioeconomic Disadvantage and Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2020 May 5;15:981-993. doi: 10.2147/COPD.S238933. eCollection 2020. PMID 32440110
- [Result] Putcha N, Fawzy A, Matsui EC, Liu MC, Bowler RP, Woodruff PG, O'Neal WK, Comellas AP, Han MK, Dransfield MT, Wells JM, Lugogo N, Gao L, Talbot CC Jr, Hoffman EA, Cooper CB, Paulin LM, Kanner RE, Criner G, Ortega VE, Barr RG, Krishnan JA, Martinez FJ, Drummond MB, Wise RA, Diette GB, Hersh CP, Hansel NN. Clinical Phenotypes of Atopy and Asthma in COPD: A Meta-analysis of SPIROMICS and COPDGene. Chest. 2020 Dec;158(6):2333-2345. doi: 10.1016/j.chest.2020.04.069. Epub 2020 May 23. PMID 32450244
- [Result] Opron K, Begley LA, Erb-Downward JR, Freeman C, Madapoosi S, Alexis NE, Barjaktarevic I, Graham Barr R, Bleecker ER, Bowler RP, Christenson SA, Comellas AP, Cooper CB, Couper DJ, Doerschuk CM, Dransfield MT, Han MK, Hansel NN, Hastie AT, Hoffman EA, Kaner RJ, Krishnan J, O'Neal WK, Ortega VE, Paine R 3rd, Peters SP, Michael Wells J, Woodruff PG, Martinez FJ, Curtis JL, Huffnagle GB, Huang YJ. Lung microbiota associations with clinical features of COPD in the SPIROMICS cohort. NPJ Biofilms Microbiomes. 2021 Feb 5;7(1):14. doi: 10.1038/s41522-021-00185-9. PMID 33547327
- [Result] Li F, Choi J, Zou C, Newell JD Jr, Comellas AP, Lee CH, Ko H, Barr RG, Bleecker ER, Cooper CB, Abtin F, Barjaktarevic I, Couper D, Han M, Hansel NN, Kanner RE, Paine R 3rd, Kazerooni EA, Martinez FJ, O'Neal W, Rennard SI, Smith BM, Woodruff PG, Hoffman EA, Lin CL. Latent traits of lung tissue patterns in former smokers derived by dual channel deep learning in computed tomography images. Sci Rep. 2021 Mar 1;11(1):4916. doi: 10.1038/s41598-021-84547-5. PMID 33649381
- [Result] Gillenwater LA, Kechris KJ, Pratte KA, Reisdorph N, Petrache I, Labaki WW, O'Neal W, Krishnan JA, Ortega VE, DeMeo DL, Bowler RP. Metabolomic Profiling Reveals Sex Specific Associations with Chronic Obstructive Pulmonary Disease and Emphysema. Metabolites. 2021 Mar 11;11(3):161. doi: 10.3390/metabo11030161. PMID 33799786
- [Result] Turnier L, Eakin M, Woo H, Dransfield M, Parekh T, Krishnan JA, Kanner R, Cooper CB, Woodruff PG, Wise R, Han MK, Romero K, Paulin LM, Peters S, Drummond B, Bleecker ER, Bowler R, Comellas AP, Couper D, Paine R, Martinez F, Barr G, Putcha N, Hansel NN. The influence of social support on COPD outcomes mediated by depression. PLoS One. 2021 Mar 17;16(3):e0245478. doi: 10.1371/journal.pone.0245478. eCollection 2021. PMID 33730034
- [Result] Kasela S, Ortega VE, Martorella M, Garudadri S, Nguyen J, Ampleford E, Pasanen A, Nerella S, Buschur KL, Barjaktarevic IZ, Barr RG, Bleecker ER, Bowler RP, Comellas AP, Cooper CB, Couper DJ, Criner GJ, Curtis JL, Han MK, Hansel NN, Hoffman EA, Kaner RJ, Krishnan JA, Martinez FJ, McDonald MN, Meyers DA, Paine R 3rd, Peters SP, Castro M, Denlinger LC, Erzurum SC, Fahy JV, Israel E, Jarjour NN, Levy BD, Li X, Moore WC, Wenzel SE, Zein J; NHLBI SubPopulations and InteRmediate Outcome Measures In COPD Study (SPIROMICS); NHLBI Trans-Omics for Precision Medicine (TOPMed) Consortium; Langelier C, Woodruff PG, Lappalainen T, Christenson SA. Genetic and non-genetic factors affecting the expression of COVID-19-relevant genes in the large airway epithelium. Genome Med. 2021 Apr 21;13(1):66. doi: 10.1186/s13073-021-00866-2. PMID 33883027
- [Result] Zhang WZ, Hoffman KL, Schiffer KT, Oromendia C, Rice MC, Barjaktarevic I, Peters SP, Putcha N, Bowler RP, Wells JM, Couper DJ, Labaki WW, Curtis JL, Han MK, Paine R 3rd, Woodruff PG, Criner GJ, Hansel NN, Diaz I, Ballman KV, Nakahira K, Choi ME, Martinez FJ, Choi AMK, Cloonan SM. Association of plasma mitochondrial DNA with COPD severity and progression in the SPIROMICS cohort. Respir Res. 2021 Apr 26;22(1):126. doi: 10.1186/s12931-021-01707-x. PMID 33902556
- [Result] Burkes RM, Couper DJ, Barjaktarevic IZ, Cooper CB, Labaki WW, Han MK, Woodruff PG, Lazarus SC, Parekh TM, Paine R 3rd, Comellas AP, Bowler RP, Loehr LR, Putcha N, Wise RA, Brown TT, Drummond MB. Age-Dependent Associations Between 25-Hydroxy Vitamin D Levels and COPD Symptoms: Analysis of SPIROMICS. Chronic Obstr Pulm Dis. 2021 Apr 27;8(2):277-291. doi: 10.15326/jcopdf.2020.0180. PMID 33829714
- [Result] Moughames E, Woo H, Galiatsatos P, Romero-Rivero K, Raju S, Tejwani V, Hoffman EA, Comellas AP, Ortega VE, Parekh T, Krishnan JA, Drummond MB, Couper D, Buhr RG, Paine R, Kaufman JD, Paulin LM, Putcha N, Hansel NN. Disparities in access to food and chronic obstructive pulmonary disease (COPD)-related outcomes: a cross-sectional analysis. BMC Pulm Med. 2021 Apr 27;21(1):139. doi: 10.1186/s12890-021-01485-8. PMID 33906617
- [Result] Pratte KA, Curtis JL, Kechris K, Couper D, Cho MH, Silverman EK, DeMeo DL, Sciurba FC, Zhang Y, Ortega VE, O'Neal WK, Gillenwater LA, Lynch DA, Hoffman EA, Newell JD Jr, Comellas AP, Castaldi PJ, Miller BE, Pouwels SD, Hacken NHTT, Bischoff R, Klont F, Woodruff PG, Paine R, Barr RG, Hoidal J, Doerschuk CM, Charbonnier JP, Sung R, Locantore N, Yonchuk JG, Jacobson S, Tal-Singer R, Merrill D, Bowler RP. Soluble receptor for advanced glycation end products (sRAGE) as a biomarker of COPD. Respir Res. 2021 Apr 27;22(1):127. doi: 10.1186/s12931-021-01686-z. PMID 33906653
- [Result] Zou C, Li F, Choi J, Haghighi B, Choi S, Rajaraman PK, Comellas AP, Newell JD, Lee CH, Barr RG, Bleecker E, Cooper CB, Couper D, Han M, Hansel NN, Kanner RE, Kazerooni EA, Kleerup EC, Martinez FJ, O'Neal W, Paine R 3rd, Rennard SI, Smith BM, Woodruff PG, Hoffman EA, Lin CL. Longitudinal Imaging-Based Clusters in Former Smokers of the COPD Cohort Associate with Clinical Characteristics: The SubPopulations and Intermediate Outcome Measures in COPD Study (SPIROMICS). Int J Chron Obstruct Pulmon Dis. 2021 May 31;16:1477-1496. doi: 10.2147/COPD.S301466. eCollection 2021. PMID 34103907
- [Result] Fawzy A, Woo H, Balasubramanian A, Barjaktarevic I, Barr RG, Bowler RP, Comellas AP, Cooper CB, Couper D, Criner GJ, Dransfield MT, Han MK, Hoffman EA, Kanner RE, Krishnan JA, Martinez FJ, McCormack M, Paine Iii R, Peters S, Wise R, Woodruff PG, Hansel NN, Putcha N. Polycythemia is Associated with Lower Incidence of Severe COPD Exacerbations in the SPIROMICS Study. Chronic Obstr Pulm Dis. 2021 Jul 28;8(3):326-335. doi: 10.15326/jcopdf.2021.0216. PMID 34197703
- [Result] O'Toole J, Woo H, Putcha N, Cooper CB, Woodruff P, Kanner RE, Paine R, Bowler RP, Comellas A, Hoth KF, Krishnan JA, Han M, Dransfield M, Iyer AS, Couper D, Peters SP, Criner G, Kim V, Barr RG, Martinez FJ, Hansel NN, Eakin MN; SPIROMICS Investigators. Comparative Impact of Depressive Symptoms and FEV1% on Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2022 Feb;19(2):171-178. doi: 10.1513/AnnalsATS.202009-1187OC. PMID 34410883
- [Result] Woo H, Brigham EP, Allbright K, Ejike C, Galiatsatos P, Jones MR, Oates GR, Krishnan JA, Cooper CB, Kanner RE, Bowler RP, Hoffman EA, Comellas AP, Criner G, Barr RG, Martinez FJ, Han M, Ortega VE, Parekh TM, Christenson S, Belz D, Raju S, Gassett A, Paulin LM, Putcha N, Kaufman JD, Hansel NN. Racial Segregation and Respiratory Outcomes among Urban Black Residents with and at Risk of Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2021 Sep 1;204(5):536-545. doi: 10.1164/rccm.202009-3721OC. PMID 33971109
- [Result] Oh AL, Mularski RA, Barjaktarevic I, Barr RG, Bowler RP, Comellas AP, Cooper CB, Criner GJ, Han MK, Hansel NN, Hoffman EA, Kanner RE, Krishnan JA, Paine R 3rd, Parekh TM, Peters SP, Christenson SA, Woodruff PG; SPIROMICS Smoking Resilience Group. Defining Resilience to Smoking-related Lung Disease: A Modified Delphi Approach from SPIROMICS. Ann Am Thorac Soc. 2021 Nov;18(11):1822-1831. doi: 10.1513/AnnalsATS.202006-757OC. PMID 33631079
- [Result] Radicioni G, Ceppe A, Ford AA, Alexis NE, Barr RG, Bleecker ER, Christenson SA, Cooper CB, Han MK, Hansel NN, Hastie AT, Hoffman EA, Kanner RE, Martinez FJ, Ozkan E, Paine R 3rd, Woodruff PG, O'Neal WK, Boucher RC, Kesimer M. Airway mucin MUC5AC and MUC5B concentrations and the initiation and progression of chronic obstructive pulmonary disease: an analysis of the SPIROMICS cohort. Lancet Respir Med. 2021 Nov;9(11):1241-1254. doi: 10.1016/S2213-2600(21)00079-5. Epub 2021 May 28. PMID 34058148
- [Result] Yee N, Markovic D, Buhr RG, Fortis S, Arjomandi M, Couper D, Anderson WH, Paine R 3rd, Woodruff PG, Han MK, Martinez FJ, Barr RG, Wells JM, Ortega VE, Hoffman EA, Kim V, Drummond MB, Bowler RP, Curtis JL, Cooper CB, Tashkin DP, Barjaktarevic IZ. Significance of FEV3/FEV6 in Recognition of Early Airway Disease in Smokers at Risk of Development of COPD: Analysis of the SPIROMICS Cohort. Chest. 2022 Apr;161(4):949-959. doi: 10.1016/j.chest.2021.10.046. Epub 2021 Nov 10. PMID 34767825
- [Result] Lakshman Kumar P, Wilson AC, Rocco A, Cho MH, Wan E, Hobbs BD, Washko GR, Ortega VE, Christenson SA, Li X, Wells JM, Bhatt SP, DeMeo DL, Lutz SM, Rossiter H, Casaburi R, Rennard SI, Lomas DA, Labaki WW, Tal-Singer R, Bowler RP, Hersh CP, Tiwari HK, Dransfield M, Thalacker-Mercer A, Meyers DA, Silverman EK, McDonald MN; COPDGene, ECLIPSE and SPIROMICS investigators. Genetic variation in genes regulating skeletal muscle regeneration and tissue remodelling associated with weight loss in chronic obstructive pulmonary disease. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1803-1817. doi: 10.1002/jcsm.12782. Epub 2021 Sep 15. PMID 34523824
- [Result] Iyer AS, Parekh TM, O'Toole J, Bhatt SP, Eakin MN, Krishnan JA, Yohannes AM, Woodruff PG, Cooper CB, Kanner RE, Hanania NA, Dransfield MT, Regan EA, Hoth KF, Kim V; COPDGene and SPIROMICS Investigators. Clinically Significant and Comorbid Anxiety and Depression Symptoms Predict Severe Respiratory Exacerbations in Smokers: A Post Hoc Analysis of the COPDGene and SPIROMICS Cohorts. Ann Am Thorac Soc. 2022 Jan;19(1):143-146. doi: 10.1513/AnnalsATS.202103-240RL. No abstract available. PMID 34343034
- [Result] Sowho MO, Koch AL, Putcha N, Woo H, Gassett A, Paulin LM, Koehler K, Barr RG, Comellas AP, Cooper CB, Barjaktarevic I, Zeidler MR, Billings ME, Bowler RP, Han MK, Kim V, Paine Iii R, Parekh TM, Krishnan JA, Peters SP, Woodruff PG, Baugh AM, Kaufman JD, Couper D, Hansel NN. Ambient Air Pollution Exposure and Sleep Quality in COPD. Chronic Obstr Pulm Dis. 2023 Jan 25;10(1):102-111. doi: 10.15326/jcopdf.2022.0350. PMID 36599095
- [Result] Pan Y, Wang D, Chaudhary MFA, Shao W, Gerard SE, Durumeric OC, Bhatt SP, Barr RG, Hoffman EA, Reinhardt JM, Christensen GE. Robust Measures of Image-Registration-Derived Lung Biomechanics in SPIROMICS. J Imaging. 2022 Nov 16;8(11):309. doi: 10.3390/jimaging8110309. PMID 36422058
- [Result] Tejwani V, Woo H, Liu C, Tillery AK, Gassett AJ, Kanner RE, Hoffman EA, Martinez FJ, Woodruff PG, Barr RG, Fawzy A, Koehler K, Curtis JL, Freeman CM, Cooper CB, Comellas AP, Pirozzi C, Paine R, Tashkin D, Krishnan JA, Sack C, Putcha N, Paulin LM, Zusman M, Kaufman JD, Alexis NE, Hansel NN. Black carbon content in airway macrophages is associated with increased severe exacerbations and worse COPD morbidity in SPIROMICS. Respir Res. 2022 Nov 14;23(1):310. doi: 10.1186/s12931-022-02225-0. PMID 36376879
- [Result] LeMaster WB, Quibrera PM, Couper D, Tashkin DP, Bleecker ER, Doerschuk CM, Ortega VE, Cooper C, Han MK, Woodruff PG, O'Neal WK, Anderson WH, Alexis NE, Bowler RP, Barr RG, Kaner RJ, Dransfield MT, Paine R 3rd, Kim V, Curtis JL, Martinez FJ, Hastie AT, Barjaktarevic I. Clinical Implications of Low Absolute Blood Eosinophil Count in the SPIROMICS COPD Cohort. Chest. 2023 Mar;163(3):515-528. doi: 10.1016/j.chest.2022.10.029. Epub 2022 Nov 4. PMID 36343688
- [Result] Esther CR Jr, O'Neal WK, Alexis NE, Koch AL, Cooper CB, Barjaktarevic I, Raffield LM, Bowler RP, Comellas AP, Peters SP, Hastie AT, Curtis JL, Ronish B, Ortega VE, Wells JM, Halper-Stromberg E, Rennard SI, Boucher RC; SPIROMICS. Prolonged, physiologically relevant nicotine concentrations in the airways of smokers. Am J Physiol Lung Cell Mol Physiol. 2023 Jan 1;324(1):L32-L37. doi: 10.1152/ajplung.00038.2022. Epub 2022 Nov 7. PMID 36342131
- [Result] Weiss JR, Serdenes R, Madtha U, Zhao H, Kim V, Lopez-Pastrana J, Eakin MN, O'Toole J, Cooper CB, Woodruff P, Kanner RE, Krishnan JA, Iyer AS, Couper D, Morrison MF. Association Among Chronic Obstructive Pulmonary Disease Severity, Exacerbation Risk, and Anxiety and Depression Symptoms in the SPIROMICS Cohort. J Acad Consult Liaison Psychiatry. 2023 Jan-Feb;64(1):45-57. doi: 10.1016/j.jaclp.2022.07.008. Epub 2022 Aug 7. PMID 35948252
- [Result] Baugh A, Buhr RG, Quibrera P, Barjaktarevic I, Barr RG, Bowler R, Han MK, Kaufman JD, Koch AL, Krishnan J, Labaki W, Martinez FJ, Mkorombindo T, Namen A, Ortega V, Paine R, Peters SP, Schotland H, Sundar K, Zeidler MR, Hansel NN, Woodruff PG, Thakur N. Risk of COPD exacerbation is increased by poor sleep quality and modified by social adversity. Sleep. 2022 Aug 11;45(8):zsac107. doi: 10.1093/sleep/zsac107. PMID 35665826
- [Result] Godbole S, Labaki WW, Pratte KA, Hill A, Moll M, Hastie AT, Peters SP, Gregory A, Ortega VE, DeMeo D, Cho MH, Bhatt SP, Wells JM, Barjaktarevic I, Stringer KA, Comellas A, O'Neal W, Kechris K, Bowler RP. A Metabolomic Severity Score for Airflow Obstruction and Emphysema. Metabolites. 2022 Apr 19;12(5):368. doi: 10.3390/metabo12050368. PMID 35629872
- [Result] Buhr RG, Barjaktarevic IZ, Quibrera PM, Bateman LA, Bleecker ER, Couper DJ, Curtis JL, Dolezal BA, Han MK, Hansel NN, Krishnan JA, Martinez FJ, McKleroy W, Paine R 3rd, Rennard SI, Tashkin DP, Woodruff PG, Kanner RE, Cooper CB; SPIROMICS Investigators. Reversible Airflow Obstruction Predicts Future Chronic Obstructive Pulmonary Disease Development in the SPIROMICS Cohort: An Observational Cohort Study. Am J Respir Crit Care Med. 2022 Sep 1;206(5):554-562. doi: 10.1164/rccm.202201-0094OC. PMID 35549640
- [Result] Madapoosi SS, Cruickshank-Quinn C, Opron K, Erb-Downward JR, Begley LA, Li G, Barjaktarevic I, Barr RG, Comellas AP, Couper DJ, Cooper CB, Freeman CM, Han MK, Kaner RJ, Labaki W, Martinez FJ, Ortega VE, Peters SP, Paine R, Woodruff P, Curtis JL, Huffnagle GB, Stringer KA, Bowler RP, Esther CR Jr, Reisdorph N, Huang YJ; SPIROMICS Research Group. Lung Microbiota and Metabolites Collectively Associate with Clinical Outcomes in Milder Stage Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2022 Aug 15;206(4):427-439. doi: 10.1164/rccm.202110-2241OC. PMID 35536732
- [Result] Wang D, Pan Y, Durumeric OC, Reinhardt JM, Hoffman EA, Schroeder JD, Christensen GE. PLOSL: Population learning followed by one shot learning pulmonary image registration using tissue volume preserving and vesselness constraints. Med Image Anal. 2022 Jul;79:102434. doi: 10.1016/j.media.2022.102434. Epub 2022 Apr 1. PMID 35430476
- [Result] Krishnan JK, Ancy KM, Oromendia C, Hoffman KL, Easthausen I, Leidy NK, Han MK, Bowler RP, Christenson SA, Couper DJ, Criner GJ, Curtis JL, Dransfield MT, Hansel NN, Iyer AS, Paine Iii R, Peters SP, Wedzicha JA, Woodruff PG, Ballman KV, Martinez FJ; SPIROMICS Investigators. Characterizing COPD Symptom Variability in the Stable State Utilizing the Evaluating Respiratory Symptoms in COPD Instrument. Chronic Obstr Pulm Dis. 2022 Apr 29;9(2):195-208. doi: 10.15326/jcopdf.2021.0263. PMID 35403414
- [Result] Belz DC, Woo H, Putcha N, Paulin LM, Koehler K, Fawzy A, Alexis NE, Barr RG, Comellas AP, Cooper CB, Couper D, Dransfield M, Gassett AJ, Han M, Hoffman EA, Kanner RE, Krishnan JA, Martinez FJ, Paine R 3rd, Peng RD, Peters S, Pirozzi CS, Woodruff PG, Kaufman JD, Hansel NN; SPIROMICS Investigators. Ambient ozone effects on respiratory outcomes among smokers modified by neighborhood poverty: An analysis of SPIROMICS AIR. Sci Total Environ. 2022 Jul 10;829:154694. doi: 10.1016/j.scitotenv.2022.154694. Epub 2022 Mar 19. PMID 35318050
- [Result] Ronish BE, Couper DJ, Barjaktarevic IZ, Cooper CB, Kanner RE, Pirozzi CS, Kim V, Wells JM, Han MK, Woodruff PG, Ortega VE, Peters SP, Hoffman EA, Buhr RG, Dolezal BA, Tashkin DP, Liou TG, Bateman LA, Schroeder JD, Martinez FJ, Barr RG, Hansel NN, Comellas AP, Rennard SI, Arjomandi M, Paine Iii R. Forced Expiratory Flow at 25%-75% Links COPD Physiology to Emphysema and Disease Severity in the SPIROMICS Cohort. Chronic Obstr Pulm Dis. 2022 Apr 29;9(2):111-121. doi: 10.15326/jcopdf.2021.0241. PMID 35114743
- [Result] Chaudhary MFA, Hoffman EA, Guo J, Comellas AP, Newell JD Jr, Nagpal P, Fortis S, Christensen GE, Gerard SE, Pan Y, Wang D, Abtin F, Barjaktarevic IZ, Barr RG, Bhatt SP, Bodduluri S, Cooper CB, Gravens-Mueller L, Han MK, Kazerooni EA, Martinez FJ, Menchaca MG, Ortega VE, Iii RP, Schroeder JD, Woodruff PG, Reinhardt JM. Predicting severe chronic obstructive pulmonary disease exacerbations using quantitative CT: a retrospective model development and external validation study. Lancet Digit Health. 2023 Feb;5(2):e83-e92. doi: 10.1016/S2589-7500(22)00232-1. PMID 36707189
- [Result] LaFon DC, Woo H, Fedarko N, Azar A, Hill H, Tebo AE, Martins TB, Han MK, Krishnan JA, Ortega VE, Barjaktarevic I, Kaner RJ, Hastie A, O'Neal WK, Couper D, Woodruff PG, Curtis JL, Hansel NN, Nahm MH, Dransfield MT, Putcha N; SPIROMICS investigators. Reduced quantity and function of pneumococcal antibodies are associated with exacerbations of COPD in SPIROMICS. Clin Immunol. 2023 May;250:109324. doi: 10.1016/j.clim.2023.109324. Epub 2023 Apr 6. PMID 37030524
- [Result] Baugh AD, Acho M, Arhin A, Barjaktarevic I, Couper D, Criner G, Han M, Hansel N, Krishnan J, Malcolm K, Namen A, Peters S, Schotland H, Sowho M, Zeidler M, Woodruff P, Thakur N. African American race is associated with worse sleep quality in heavy smokers. J Clin Sleep Med. 2023 Aug 1;19(8):1523-1532. doi: 10.5664/jcsm.10624. PMID 37128722
- [Result] Wang JM, Labaki WW, Murray S, Martinez FJ, Curtis JL, Hoffman EA, Ram S, Bell AJ, Galban CJ, Han MK, Hatt C. Machine learning for screening of at-risk, mild and moderate COPD patients at risk of FEV1 decline: results from COPDGene and SPIROMICS. Front Physiol. 2023 Apr 21;14:1144192. doi: 10.3389/fphys.2023.1144192. eCollection 2023. PMID 37153221
- [Result] Arjomandi M, Zeng S, Chen J, Bhatt SP, Abtin F, Barjaktarevic I, Barr RG, Bleecker ER, Buhr RG, Criner GJ, Comellas AP, Couper DJ, Curtis JL, Dransfield MT, Fortis S, Han MK, Hansel NN, Hoffman EA, Hokanson JE, Kaner RJ, Kanner RE, Krishnan JA, Labaki WW, Lynch DA, Ortega VE, Peters SP, Woodruff PG, Cooper CB, Bowler RP, Paine R 3rd, Rennard SI, Tashkin DP; and the COPDGene and SPIROMICS Investigators. Changes in Lung Volumes with Spirometric Disease Progression in COPD. Chronic Obstr Pulm Dis. 2023 Jul 26;10(3):270-285. doi: 10.15326/jcopdf.2022.0363. PMID 37199719
- [Result] Izquierdo M, Marion CR, Genese F, Newell JD, O'Neal WK, Li X, Hawkins GA, Barjaktarevic I, Barr RG, Christenson S, Cooper CB, Couper D, Curtis J, Han MK, Hansel NN, Kanner RE, Martinez FJ, Paine R 3rd, Tejwani V, Woodruff PG, Zein JG, Hoffman EA, Peters SP, Meyers DA, Bleecker ER, Ortega VE; SubPopulations and InteRmediate Outcome Measures In COPD Study (SPIROMICS) investigators. Impact of Bronchiectasis on COPD Severity and Alpha-1 Antitrypsin Deficiency as a Risk Factor in Individuals with a Heavy Smoking History. Chronic Obstr Pulm Dis. 2023 Jul 26;10(3):199-210. doi: 10.15326/jcopdf.2023.0388. PMID 37199731
- [Result] Barjaktarevic I, Cooper CB, Shing T, Buhr RG, Hoffman EA, Woodruff PG, Drummond MB, Kanner RE, Han MK, Hansel NN, Bowler RP, Kinney GL, Jacobson S, Morris MA, Martinez FJ, Ohar J, Couper D, Tashkin DP. Impact of Marijuana Smoking on COPD Progression in a Cohort of Middle-Aged and Older Persons. Chronic Obstr Pulm Dis. 2023 Jul 26;10(3):234-247. doi: 10.15326/jcopdf.2022.0378. PMID 37199732
- [Result] DiLillo KM, Norman KC, Freeman CM, Christenson SA, Alexis NE, Anderson WH, Barjaktarevic IZ, Barr RG, Comellas AP, Bleecker ER, Boucher RC, Couper DJ, Criner GJ, Doerschuk CM, Wells JM, Han MK, Hoffman EA, Hansel NN, Hastie AT, Kaner RJ, Krishnan JA, Labaki WW, Martinez FJ, Meyers DA, O'Neal WK, Ortega VE, Paine R 3rd, Peters SP, Woodruff PG, Cooper CB, Bowler RP, Curtis JL, Arnold KB; SPIROMICS investigators. A blood and bronchoalveolar lavage protein signature of rapid FEV1 decline in smoking-associated COPD. Sci Rep. 2023 May 22;13(1):8228. doi: 10.1038/s41598-023-32216-0. PMID 37217548
- [Result] Angelini ED, Yang J, Balte PP, Hoffman EA, Manichaikul AW, Sun Y, Shen W, Austin JHM, Allen NB, Bleecker ER, Bowler R, Cho MH, Cooper CS, Couper D, Dransfield MT, Garcia CK, Han MK, Hansel NN, Hughes E, Jacobs DR, Kasela S, Kaufman JD, Kim JS, Lappalainen T, Lima J, Malinsky D, Martinez FJ, Oelsner EC, Ortega VE, Paine R, Post W, Pottinger TD, Prince MR, Rich SS, Silverman EK, Smith BM, Swift AJ, Watson KE, Woodruff PG, Laine AF, Barr RG. Pulmonary emphysema subtypes defined by unsupervised machine learning on CT scans. Thorax. 2023 Nov;78(11):1067-1079. doi: 10.1136/thorax-2022-219158. Epub 2023 Jun 2. PMID 37268414
- [Result] Ryu MH, Yun JH, Morrow JD, Saferali A, Castaldi P, Chase R, Stav M, Xu Z, Barjaktarevic I, Han M, Labaki W, Huang YJ, Christenson S, O'Neal W, Bowler R, Sin DD, Freeman CM, Curtis JL, Hersh CP. Blood Gene Expression and Immune Cell Subtypes Associated with Chronic Obstructive Pulmonary Disease Exacerbations. Am J Respir Crit Care Med. 2023 Aug 1;208(3):247-255. doi: 10.1164/rccm.202301-0085OC. PMID 37286295
- [Result] Hill AC, Guo C, Litkowski EM, Manichaikul AW, Yu B, Konigsberg IR, Gorbet BA, Lange LA, Pratte KA, Kechris KJ, DeCamp M, Coors M, Ortega VE, Rich SS, Rotter JI, Gerzsten RE, Clish CB, Curtis JL, Hu X, Obeidat ME, Morris M, Loureiro J, Ngo D, O'Neal WK, Meyers DA, Bleecker ER, Hobbs BD, Cho MH, Banaei-Kashani F, Bowler RP. Large scale proteomic studies create novel privacy considerations. Sci Rep. 2023 Jun 7;13(1):9254. doi: 10.1038/s41598-023-34866-6. PMID 37286633
- [Result] Van Buren E, Radicioni G, Lester S, O'Neal WK, Dang H, Kasela S, Garudadri S, Curtis JL, Han MK, Krishnan JA, Wan ES, Silverman EK, Hastie A, Ortega VE, Lappalainen T, Nawijn MC, Berge MVD, Christenson SA, Li Y, Cho MH, Kesimer M, Kelada SNP. Genetic regulators of sputum mucin concentration and their associations with COPD phenotypes. PLoS Genet. 2023 Jun 23;19(6):e1010445. doi: 10.1371/journal.pgen.1010445. eCollection 2023 Jun. PMID 37352370
- [Result] Motahari A, Barr RG, Han MK, Anderson WH, Barjaktarevic I, Bleecker ER, Comellas AP, Cooper CB, Couper DJ, Hansel NN, Kanner RE, Kazerooni EA, Lynch DA, Martinez FJ, Newell JD Jr, Schroeder JD, Smith BM, Woodruff PG, Hoffman EA; SPIROMICS Group. Repeatability of Pulmonary Quantitative Computed Tomography Measurements in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2023 Sep 15;208(6):657-665. doi: 10.1164/rccm.202209-1698PP. No abstract available. PMID 37490608
- [Result] Hansel NN, Woo H, Koehler K, Gassett A, Paulin LM, Alexis NE, Putcha N, Lorizio W, Fawzy A, Belz D, Sack C, Barr RG, Martinez FJ, Han MK, Woodruff P, Pirozzi C, Paine R 3rd, Barjaktarevic I, Cooper CB, Ortega V, Zusman M, Kaufman JD. Indoor Pollution and Lung Function Decline in Current and Former Smokers: SPIROMICS AIR. Am J Respir Crit Care Med. 2023 Nov 15;208(10):1042-1051. doi: 10.1164/rccm.202302-0207OC. PMID 37523421
- [Result] McKleroy W, Shing T, Anderson WH, Arjomandi M, Awan HA, Barjaktarevic I, Barr RG, Bleecker ER, Boscardin J, Bowler RP, Buhr RG, Criner GJ, Comellas AP, Curtis JL, Dransfield M, Doerschuk CM, Dolezal BA, Drummond MB, Han MK, Hansel NN, Helton K, Hoffman EA, Kaner RJ, Kanner RE, Krishnan JA, Lazarus SC, Martinez FJ, Ohar J, Ortega VE, Paine R 3rd, Peters SP, Reinhardt JM, Rennard S, Smith BM, Tashkin DP, Couper D, Cooper CB, Woodruff PG. Longitudinal Follow-Up of Participants With Tobacco Exposure and Preserved Spirometry. JAMA. 2023 Aug 1;330(5):442-453. doi: 10.1001/jama.2023.11676. PMID 37526720
- [Result] Wendt CH, Bowler RP, Demorest C, Hastie A, Labaki WW, Chen M, Carmella SG, Hecht SS. Levels of Urinary Mercapturic Acids of Acrolein, Methacrolein, Crotonaldehyde, and Methyl Vinyl Ketone in Relationship to Chronic Obstructive Pulmonary Disease in Cigarette Smokers of the Subpopulations and Intermediate Outcome Measures in COPD Study (SPIROMICS). Chem Res Toxicol. 2023 Sep 19. doi: 10.1021/acs.chemrestox.3c00197. Online ahead of print. PMID 37725788
- [Result] Koch AL, Shing TL, Namen A, Couper D, Smith B, Barr RG, Bhatt S, Putcha N, Baugh A, Saha AK, Ziedler M, Comellas A, Cooper CB, Barjaktarevic I, Bowler RP, Han MK, Kim V, Paine R 3rd, Kanner RE, Krishnan JA, Martinez FJ, Woodruff PG, Hansel NN, Hoffman EA, Peters SP, Ortega VE; SubPopulations and InteRmediate Outcome Measures in COPD Study (SPIROMICS) Investigators. Lung Structure and Risk of Sleep Apnea in SPIROMICS. Chronic Obstr Pulm Dis. 2024 Jan 25;11(1):26-36. doi: 10.15326/jcopdf.2023.0411. PMID 37931592
- [Derived] Awan HA, Chaudhary MFA, El-Sokkary AD, Hoffman EA, Comellas AP, Guo J, Barjaktarevic IZ, Barr RG, Bhatt SP, Bodduluri S, Bowler RP, Vargas Buonfiglio LG, Cooper CB, Fawzy A, Hastie AT, Labaki WW, Martinez FJ, Menchaca MG, O'Neal W, Paine R 3rd, Schroeder JD, Woodruff PG, Curtis JL, Reinhardt JM. Association of Lung Quantitative CT Scan Textures With Systemic Inflammation and Mortality in COPD. Chest. 2025 Nov;168(5):1107-1119. doi: 10.1016/j.chest.2025.04.017. Epub 2025 Apr 22. PMID 40268239
- [Derived] Zhang X, Cooper CB, Prince MR, Ambale-Venkatesh B, Agarwal PP, Backman MC, Bluemke DA, Couper D, Dashnaw SM, Finn JP, Hansel NN, Hoffman EA, Jambawalikar S, Kitzman DW, Krishnan JA, Lee YJ, Lima JAC, Liu J, Menchaca MG, Ohar J, Ortega VE, Paine R 3rd, Peters SP, Schroeder JD, Vogel-Claussen J, Woodruff PG, Barr RG, Shen W. MRI-assessed Dynamic Hyperinflation Induced by Tachypnea in Chronic Obstructive Pulmonary Disease: The SPIROMICS-HF Study. Radiol Cardiothorac Imaging. 2025 Feb;7(1):e240053. doi: 10.1148/ryct.240053. PMID 39836055
- [Derived] Yang H, Yang Y, Wang F, Miao C, Chen Z, Zha S, Li X, Chen J, Song A, Chen R, Liang Z. Clinical and Prognostic Differences in Mild to Moderate COPD With and Without Emphysema. Chest. 2025 Mar;167(3):724-735. doi: 10.1016/j.chest.2024.10.020. Epub 2024 Oct 23. PMID 39454999
- [Derived] Bell AJ, Ram S, Labaki WW, Murray S, Kazerooni EA, Galban S, Martinez FJ, Hatt CR, Wang JM, Ivanov V, McGettigan P, Khokhlovich E, Maiorino E, Suryadevara R, Boueiz A, Castaldi PJ, Mirkes EM, Zinovyev A, Gorban AN, Galban CJ, Han MK. Temporal Exploration of Chronic Obstructive Pulmonary Disease Phenotypes: Insights from the COPDGene and SPIROMICS Cohorts. Am J Respir Crit Care Med. 2025 Apr;211(4):569-576. doi: 10.1164/rccm.202401-0127OC. PMID 39269427
- [Derived] Suri R, Markovic D, Woo H, Arjomandi M, Barr RG, Bowler RP, Criner G, Curtis JL, Dransfield MT, Drummond MB, Fortis S, Han MK, Hoffman EA, Kaner RJ, Kaufman JD, Krishnan JA, Martinez FJ, Ohar J, Ortega VE, Paine R 3rd, Soler X, Woodruff PG, Hansel NN, Cooper CB, Tashkin DP, Buhr RG, Barjaktarevic IZ. The Effect of Chronic Altitude Exposure on Chronic Obstructive Pulmonary Disease Outcomes in the SPIROMICS Cohort: An Observational Cohort Study. Am J Respir Crit Care Med. 2024 Nov 15;210(10):1210-1218. doi: 10.1164/rccm.202310-1965OC. PMID 38507607
- [Derived] Barjaktarevic I, Cooper CB, Shing T, Buhr RG, Hoffman EA, Woodruff PG, Drummond MB, Kanner RE, Han MK, Hansel NN, Bowler RP, Kinney GL, Jacobson S, Morris MA, Martinez FJ, Ohar J, Couper D, Tashkin DP. Effect of marijuana smoking on lung function change in older ever tobacco smokers. Eur Respir J. 2022 Sep 22;60(3):2201133. doi: 10.1183/13993003.01133-2022. Print 2022 Sep. No abstract available. PMID 36137583
- [Derived] Baugh AD, Shiboski S, Hansel NN, Ortega V, Barjaktarevic I, Barr RG, Bowler R, Comellas AP, Cooper CB, Couper D, Criner G, Curtis JL, Dransfield M, Ejike C, Han MK, Hoffman E, Krishnan J, Krishnan JA, Mannino D, Paine R 3rd, Parekh T, Peters S, Putcha N, Rennard S, Thakur N, Woodruff PG. Reconsidering the Utility of Race-Specific Lung Function Prediction Equations. Am J Respir Crit Care Med. 2022 Apr 1;205(7):819-829. doi: 10.1164/rccm.202105-1246OC. PMID 34913855
- [Derived] Esther CR Jr, O'Neal WK, Anderson WH, Kesimer M, Ceppe A, Doerschuk CM, Alexis NE, Hastie AT, Barr RG, Bowler RP, Wells JM, Oelsner EC, Comellas AP, Tesfaigzi Y, Kim V, Paulin LM, Cooper CB, Han MK, Huang YJ, Labaki WW, Curtis JL, Boucher RC; Subpopulations and Intermediate Outcome Measures in COPD Study. Identification of Sputum Biomarkers Predictive of Pulmonary Exacerbations in COPD. Chest. 2022 May;161(5):1239-1249. doi: 10.1016/j.chest.2021.10.049. Epub 2021 Nov 18. PMID 34801592
- [Derived] Fortis S, Comellas AP, Bhatt SP, Hoffman EA, Han MK, Bhakta NR, Paine R 3rd, Ronish B, Kanner RE, Dransfield M, Hoesterey D, Buhr RG, Barr RG, Dolezal B, Ortega VE, Drummond MB, Arjomandi M, Kaner RJ, Kim V, Curtis JL, Bowler RP, Martinez F, Labaki WW, Cooper CB, O'Neal WK, Criner G, Hansel NN, Krishnan JA, Woodruff P, Couper D, Tashkin D, Barjaktarevic I. Ratio of FEV1/Slow Vital Capacity of < 0.7 Is Associated With Clinical, Functional, and Radiologic Features of Obstructive Lung Disease in Smokers With Preserved Lung Function. Chest. 2021 Jul;160(1):94-103. doi: 10.1016/j.chest.2021.01.067. Epub 2021 Feb 1. PMID 33539837
- [Derived] Dunican EM, Elicker BM, Henry T, Gierada DS, Schiebler ML, Anderson W, Barjaktarevic I, Barr RG, Bleecker ER, Boucher RC, Bowler R, Christenson SA, Comellas A, Cooper CB, Couper D, Criner GJ, Dransfield M, Doerschuk CM, Drummond MB, Hansel NN, Han MK, Hastie AT, Hoffman EA, Krishnan JA, Lazarus SC, Martinez FJ, McCulloch CE, O'Neal WK, Ortega VE, Paine R 3rd, Peters S, Schroeder JD, Woodruff PG, Fahy JV. Mucus Plugs and Emphysema in the Pathophysiology of Airflow Obstruction and Hypoxemia in Smokers. Am J Respir Crit Care Med. 2021 Apr 15;203(8):957-968. doi: 10.1164/rccm.202006-2248OC. PMID 33180550
- See also: Study Website — https://spiromics.org